CLINICAL TRIAL: NCT03982186
Title: A Phase 2b, Multicenter, Double-blind, Active-controlled, Randomized Study to Investigate the Efficacy and Safety of Different Combination Regimens Including JNJ-73763989 and/or JNJ-56136379 for the Treatment of Chronic Hepatitis B Virus Infection
Brief Title: A Study of Different Combination Regimens Including JNJ-73763989 and/or JNJ-56136379 for the Treatment of Chronic Hepatitis B Virus Infection
Acronym: REEF-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Sciences Ireland UC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR108608; 2019-000622-22 (EudraCT Number); 73763989HPB2001 (Other: Janssen Sciences Ireland UC)
Record Dates: First submitted 2019-06-10; First posted 2019-06-11 (Actual); Results first posted 2024-07-10 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — JNJ-56136379

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- Arm 1: JNJ-73763989 (medium dose) + JNJ-56136379 + NA (Experimental): Participants will receive medium dose of JNJ-73763989 along with JNJ-56136379 and nucleos(t)ide analog (NA) treatment (either entecavir [ETV], tenofovir disoproxil fumarate [TDF], or tenofovir alafenamide [TAF]) up to 48 weeks.
  Interventions: Drug: JNJ-73763989; Drug: JNJ-56136379; Drug: Nucleos(t)ide Analog (NA)
- Arm 2: JNJ-73763989 (high dose) + Placebo + NA (Experimental): Participants will receive high dose of JNJ-73763989 along with placebo for JNJ-56136379 and NA (either ETV, TDF, or TAF) up to 48 weeks.
  Interventions: Drug: JNJ-73763989; Drug: Placebo for JNJ-56136379; Drug: Nucleos(t)ide Analog (NA)
- Arm 3: JNJ-73763989 (medium dose) + Placebo + NA (Experimental): Participants will receive medium dose of JNJ-73763989 along with placebo for JNJ-56136379 and NA (either ETV, TDF, or TAF) up to 48 weeks.
  Interventions: Drug: JNJ-73763989; Drug: Placebo for JNJ-56136379; Drug: Nucleos(t)ide Analog (NA)
- Arm 4: JNJ-73763989 (low dose) + Placebo + NA (Experimental): Participants will receive low dose of JNJ-73763989 along with placebo for JNJ-56136379 and NA (either ETV, TDF, or TAF) up to 48 weeks.
  Interventions: Drug: JNJ-73763989; Drug: Placebo for JNJ-56136379; Drug: Nucleos(t)ide Analog (NA)
- Arm 5: Placebo + JNJ-56136379 + NA (Experimental): Participants will receive placebo for JNJ-73763989 and a fixed dose of JNJ-56136379 along with NA (either ETV, TDF, or TAF) up to 48 weeks.
  Interventions: Drug: Placebo for JNJ-73763989; Drug: JNJ-56136379; Drug: Nucleos(t)ide Analog (NA)
- Arm 6 (Control): Placebo + Placebo + NA (Placebo Comparator): Participants will receive placebo for JNJ-73763989 and placebo for JNJ-56136379 along with NA (either ETV, TDF, or TAF) up to 48 weeks.
  Interventions: Drug: Placebo for JNJ-73763989; Drug: Placebo for JNJ-56136379; Drug: Nucleos(t)ide Analog (NA)

INTERVENTIONS:
Drug: JNJ-73763989 — JNJ-73763989 will be administered as medium dose (Arms 1 and 3), high dose (Arm 2), and low dose (Arm 4) as subcutaneous injection.
  Arms: Arm 1: JNJ-73763989 (medium dose) + JNJ-56136379 + NA; Arm 2: JNJ-73763989 (high dose) + Placebo + NA; Arm 3: JNJ-73763989 (medium dose) + Placebo + NA; Arm 4: JNJ-73763989 (low dose) + Placebo + NA
Drug: Placebo for JNJ-73763989 — Placebo for JNJ-73763989 will be administered as subcutaneous injection.
  Arms: Arm 5: Placebo + JNJ-56136379 + NA; Arm 6 (Control): Placebo + Placebo + NA
Drug: JNJ-56136379 — JNJ-56136379 tablets will be administered orally.
  Arms: Arm 1: JNJ-73763989 (medium dose) + JNJ-56136379 + NA; Arm 5: Placebo + JNJ-56136379 + NA
Drug: Placebo for JNJ-56136379 — Placebo for JNJ-56136379 tablets will be administered orally.
  Arms: Arm 2: JNJ-73763989 (high dose) + Placebo + NA; Arm 3: JNJ-73763989 (medium dose) + Placebo + NA; Arm 4: JNJ-73763989 (low dose) + Placebo + NA; Arm 6 (Control): Placebo + Placebo + NA
Drug: Nucleos(t)ide Analog (NA) — NA treatment that is either of ETV, TDF or TAF tablets will be administered orally.

SUMMARY:
The purpose of this study is to establish the dose-response relationship for antiviral activity of 3 dose levels of JNJ-73763989+nucleos(t)ide analog (NA) and to evaluate the efficacy of combination regimens of JNJ-73763989+NA (with and without JNJ-56136379) and of JNJ-56136379+NA.

DETAILED DESCRIPTION:
Hepatitis B virus (HBV) is a small deoxyribonucleic acid virus that specifically infects the human liver. The acute phase of infection is either followed by an immune controlled state or progresses to chronic hepatitis B. The worldwide estimated prevalence of chronic HBV infection is about 292 million people affected. Hepatitis B surface antigen (HBsAg) seroclearance is currently considered to be associated with the most thorough suppression of HBV replication (termed functional cure). With current available NA treatment strategies, rate of HBsAg seroclearance remains very low (around 3 percent [%]) even under long-term treatment. Also, with the persistently high global prevalence of HBV-associated mortality, there is a medical need for more effective finite treatment options that lead to sustained HBsAg seroclearance. JNJ-73763989 is a liver-targeted antiviral therapeutic for subcutaneous injection designed to treat chronic HBV infection via ribonucleic acid interference mechanism. JNJ-56136379 is an orally administered capsid assembly modulator that is being developed for the treatment of chronic HBV infection. The aim of the study is to evaluate efficacy as measured by proportion of participants who completed 48-week study intervention and qualified for stopping NA treatment at Week 48. The study includes: Screening phase (4 weeks), Double-blind study intervention phase (from Day 1 up to Week 48), and Follow-up phase (48 weeks after end of investigational intervention with a maximum duration of 96 weeks). The duration of individual study participation will be between 100 and 150 weeks. Safety and tolerability (including adverse events [AEs] and Serious AEs, laboratory assessments, electrocardiogram [ECG], vital signs, physical examination), efficacy (including HBsAg seroclearance), and pharmacokinetics will be assessed throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Medically stable based on physical examination, medical history, vital signs, electrocardiogram (ECG) at screening
* Chronic hepatitis B virus (HBV) infection with documentation at least 6 months prior to screening
* Hepatitis B surface antigen (HBsAg) greater than (>) 100 International Units per Milliliter (IU/mL) at screening
* Body mass index (BMI) between 18.0 and 35.0 kilogram per meter square (kg/m^2), extremes included
* Highly effective contraceptive measures in place for female participants of childbearing potential or male participants with female partners of childbearing potential
* Liver fibrosis stage 0-2 (Metavir) or Fibroscan less than (<) 9 Kilopascal (kPa) at screening

Exclusion Criteria:

* Evidence of infection with hepatitis A, C, D or E virus infection or evidence of human immunodeficiency, virus type 1 (HIV-1) or HIV-2 infection at screening
* History or evidence of clinical signs/symptoms of hepatic decompensation including but not limited to: portal hypertension, ascites, hepatic encephalopathy, esophageal varices or any laboratory abnormalities indicating a reduced liver function as defined in the protocol
* Evidence of liver disease of non-HBV etiology
* Signs of hepatocellular carcinoma (HCC)
* Significant laboratory abnormalities as defined in the protocol at screening
* Participants with a history of malignancy within 5 years before screening
* Abnormal sinus rhythm or ECG parameters at screening as defined in the protocol
* History of or current cardiac arrhythmia or history or clinical evidence of significant or unstable cardiac disease
* Participants with any current or previous illness for which, in the opinion of the investigator and/or sponsor, participation would not be in the best interest of the participant
* History of or current clinically significant skin disease or drug rash
* Participants with known allergies, hypersensitivity, or intolerance to JNJ-3989 and JNJ 6379 or their excipients or excipients of the placebo content
* Contraindications to the use of entecavir (ETV), tenofovir disoproxil fumarate (TDF), or tenofovir alafenamide (TAF) per local prescribing information
* Participants who have taken any therapies disallowed per protocol
* Female participants who are pregnant, or breast-feeding, or planning to become pregnant while enrolled in this study or within 90 days after the last dose of study intervention
* Male participants who plan to father a child while enrolled
* Participants who had or planned major surgery, (example, requiring general anesthesia) or who have received an organ transplant
* Vulnerable participants (example, incarcerated individuals, individuals under a legal protection measure)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 471 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-03-29 (Actual); Study Completion 2022-04-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Sciences Ireland UC Clinical Trial, Study Director — Janssen Sciences Ireland UC
Locations (108):
- United States (8):
  - The Office of Franco Felizarta, MD, Bakersfield, California
  - Ruane Clinical Research Group Inc, Los Angeles, California
  - Southern California GI and Liver Center, San Clemente, California
  - Johns Hopkins Office of Capital Region Research - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Johns Hopkins University, Baltimore, Maryland
  - Washington University School Of Medicine, St Louis, Missouri
  - I.D. Care, Inc., Hillsborough, New Jersey
  - NYU Hepatology Associates, New York, New York
- Belgium (5):
  - Cliniques Universitaires Saint Luc, Brussels
  - UZ Antwerpen, Edegem
  - UZA-SGS, Edegem
  - Universitair Ziekenhuis Gent, Ghent
  - UZ Leuven, Leuven
- Brazil (3):
  - Fundacao de Medicina Tropical Doutor Heitor Vieira Dourado - FMT, Manaus
  - Universidade Federal da Bahia - Hospital Professor Edgard Santos, Salvador
  - Hospital Das Clinicas Da Faculdade De Medicina Da USP, São Paulo
- Canada (5):
  - University of Calgary, Calgary, Alberta
  - University of Alberta - Faculty of Medicine & Dentistry, Edmonton, Alberta
  - GI Research Institute (G.I.R.I.), Vancouver, British Columbia
  - Vancouver ID Research and Care Centre Society, Vancouver, British Columbia
  - Toronto General Hospital, Toronto, Ontario
- Nanfang Hospital, Guangzhou, China
- Czechia (4):
  - FN Hradec Kralove, Hradec Králové
  - RESEARCH SITE s.r.o., Pilsen
  - KLIN MED s.r.o, Prague
  - IKEM, Prague
- France (8):
  - Hopital Beaujon, Clichy
  - CHU de Grenoble Hopital Albert Michallon, Grenoble
  - Hopital de La Croix Rousse, Lyon
  - Hopital Saint Joseph, Marseille
  - CHU de Nantes hotel Dieu, Nantes
  - Hopital Saint-Antoine, Paris
  - Chu Rennes Hopital Pontchaillou, Rennes
  - Hopital Paul Brousse, Villejuif
- Germany (8):
  - EPIMED GmbH, Berlin
  - Universitatsklinikum Essen, Essen
  - Universitätsklinikum Johann Wolfgang Goethe- Universität Frankfurt Medizinische Klinik 1, Frankfurt
  - ICH Study Center GmbH & Co. KG, Hamburg
  - University Medical Center, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Universitaetsklinikum Leipzig, Leipzig
  - Universitatsmedizin der Johannes Gutenberg Universitat Mainz, Mainz
- Hong Kong (2):
  - The University of Hong Kong, Hong Kong
  - The Chinese University of Hong Kong, Shatin
- Italy (5):
  - Azienda Ospedaliera Universitaria Policlinico G. Martino, Messina
  - Irccs Ospedale Maggiore Di Milano, Milan
  - Azienda Ospedaliero-Universitaria di Modena, Ospedale di Baggiovara, Modena
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - Universita degli Studi di Roma 'La Sapienza' - Umberto I Policlinico di Roma, Rome
- Japan (15):
  - Tokyo Medical and Dental University Hospital, Bunkyō City
  - Chiba University Hospital, Chiba
  - Fukui-ken Saiseikai Hospital, Fukui
  - Fukuyama City Hospital, Fukuyama
  - Hiroshima University Hospital, Hiroshima
  - Kagawa Prefectural Central Hospital, Kagawa
  - Nara Medical University Hospital, Kashihara
  - Musashino Red Cross Hospital, Musashino
  - National Hospital Organization Nagasaki Medical Center, Nagasaki
  - Nagoya City University Hospital, Nagoya
  - The Hospital of Hyogo College of Medicine, Nishinomiya
  - Hokkaido University Hospital, Sapporo
  - Osaka University Hospital, Suita-shi
  - Toranomon Hospital, Tokyo
  - Fujita Health University Hospital, Toyoake
- Malaysia (4):
  - Hospital Sultanah Bahiyah, Alor Star
  - Hospital Selayang, Batu Caves
  - Hospital University Sains Malaysia, Kota Bharu
  - University Malaya Medical Centre, Kuala Lumpur
- Poland (5):
  - Wojewodzki Szpital Obserwacyjno-Zakazny im. Tadeusza Browicza w Bydgoszczy, Bydgoszcz
  - Neutrum Lekarze M.Hlebowicz i Partnerzy spolka partnerska, Gdansk
  - ID Clinic, Mysłowice
  - Wojewodzki Szpital Zakazny w Warszawie, Warsaw
  - SP ZOZ Wroclawskie Centrum Zdrowia, Wroclaw
- Russia (11):
  - Ural State Medical University, Chelyabinsk
  - Krasnoyarsk Regional Center For AIDS And Infectious Diseases Treatment And Prophylaxis, Krasnoyarsk
  - Clinic of the Modern Medicine, Moscow
  - Medical Center SibNovoMed LLC, Novosibirsk
  - St. Petersburg City Center for AIDS and Infectious Diseases Treatment and Prophylaxis, Saint Petersburg
  - Clinical Infectious Diseases Hospital n. a. S.P. Botkin, Saint Petersburg
  - Republican Clinical Infectious Hospital, Saint Petersburg
  - Medical Company Hepatolog Ltd, Samara
  - Smolensk Regional Clinical Hospital, Smolensk
  - Stavropol State Medical University, Stavropol
  - Sverdlovsk Regional Clinical Hospital #1, Yekaterinburg
- South Korea (4):
  - Seoul National University Hospital, Seoul
  - Severance Hospital Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (6):
  - Hosp Clinic de Barcelona, Barcelona
  - Hosp Univ Vall D Hebron, Barcelona
  - Hosp. Univ. 12 de Octubre, Madrid
  - Hospital Puerta De Hierro, Madrid
  - Hosp. Univ. Marques de Valdecilla, Santander
  - Hosp. Gral. Univ. Valencia, Valencia
- Thailand (4):
  - King Chulalongkorn Memorial Hospital, Bangkok
  - Siriraj Hospital, Bangkok
  - Chiang Mai University Hospital, Chiang Mai
  - Prince Of Songkla University, Songkhla
- Turkey (Türkiye) (6):
  - Hacettepe University Hospital, Ankara
  - Ankara University Medical Faculty, Ankara
  - Ankara Bilkent Sehir Hastanesi, Ankara
  - Istanbul University Cerrahpasa Medical Faculty, Istanbul
  - Ege University Medical of Faculty, Department of Gastroenterology, Izmir
  - Karadeniz Teknik University Medical Faculty, Trabzon
- United Kingdom (4):
  - NHS Greater Glasgow and Clyde - Gartnavel General Hospital, Glasgow
  - Grahame Hayton Unit, London
  - Kings College Hospital, London
  - St Georges University of London and St George's University Hospitals NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

REFERENCES:
- [Derived] Verbinnen T, Lathouwers E, Jezorwski J, Biermer M, Augustyns I, Grant C, Agarwal K, Yuen MF, De Meyer S, Lenz O. Viral sequence analysis of chronic hepatitis B patients treated with the siRNA JNJ-73763989 in phase II clinical trials. JHEP Rep. 2025 Oct 9;7(12):101618. doi: 10.1016/j.jhepr.2025.101618. eCollection 2025 Dec. PMID 41362713
- [Derived] Yuen MF, Asselah T, Jacobson IM, Brunetto MR, Janssen HLA, Takehara T, Hou JL, Kakuda TN, Lambrecht T, Beumont M, Kalmeijer R, Guinard-Azadian C, Mayer C, Jezorwski J, Verbinnen T, Lenz O, Shukla U, Biermer M; REEF-1 Study Group. Efficacy and safety of the siRNA JNJ-73763989 and the capsid assembly modulator JNJ-56136379 (bersacapavir) with nucleos(t)ide analogues for the treatment of chronic hepatitis B virus infection (REEF-1): a multicentre, double-blind, active-controlled, randomised, phase 2b trial. Lancet Gastroenterol Hepatol. 2023 Sep;8(9):790-802. doi: 10.1016/S2468-1253(23)00148-6. Epub 2023 Jul 10. PMID 37442152

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: JNJ-73763989 100 mg + JNJ-56136379 250 mg + NA: Participants with chronic hepatitis B (CHB) received JNJ-73763989 100 milligrams (mg) as subcutaneous (SC) injection once every 4 weeks along with JNJ-56136379 250 mg as oral tablet once daily and Nucleos(t)ide Analog (NA) (either entecavir [ETV] monohydrate 0.5 mg, tenofovir disoproxil fumarate [TDF] 300 mg, or tenofovir alafenamide [TAF] 25 mg) tablet orally once daily up to 48 weeks during double blind phase. Participants who met NA treatment completion criteria at Week 48 that is alanine aminotransferase (ALT) less than (<) 3*upper limit of normal (ULN), hepatitis B virus (HBV) deoxyribonucleic acid (DNA) < lower limit of quantification (LLOQ), hepatitis B e antigen (HBeAg) negative, hepatitis B surface antigen (HBsAg) less than (<) 10 international unit per milliliter (IU/mL) entered follow up phase 1: participants who did not meet NA treatment completion criteria or did not stop NA, follow up phase 2: participants who Met NA treatment completion criteria at Week 44 and stopped NA at Week 48, follow up phase 3: participants who met NA treatment completion criteria after Week 44 and stopped NA during follow-up and were monitored closely for 48 weeks. Participants who did not meet above criteria at Week 48 continued NA treatment during 48-week follow-up phase. Participants who completed NA treatment during the follow-up phase entered the extended follow up phase up to 48 weeks (extended follow up Week 1 to extended follow up Week 48).
- Arm 2: JNJ-73763989 200 mg + Placebo + NA: Participants with CHB received JNJ-73763989 200 mg as SC injection once every 4 weeks along with placebo matching to JNJ-56136379 tablet orally once daily and NA (either ETV 0.5 mg, TDF 300 mg, or TAF 25 mg) tablet orally once daily up to 48 weeks during double blind phase. Participants who met NA treatment completion criteria at Week 48 that is ALT <3*ULN, HBV DNA < LLOQ, HBeAg negative, HBsAg <10 IU/mL entered follow up phase 1: participants who did not meet NA treatment completion criteria or did not stop NA, follow up phase 2: participants who Met NA treatment completion criteria at Week 44 and stopped NA at Week 48, follow up phase 3: participants who met NA treatment completion criteria after Week 44 and stopped NA during follow-up and were monitored closely for 48 weeks. Participants who did not meet above criteria at Week 48 continued NA treatment during 48-week follow-up phase. Participants who completed NA treatment during the follow-up phase entered the extended follow up phase up to 48 weeks (extended follow up Week 1 to extended follow up Week 48).
- Arm 3: JNJ-73763989 100 mg + Placebo + NA: Participants with CHB received JNJ-73763989 100 mg as SC injection once every 4 weeks along with placebo matching to JNJ-56136379 tablet orally once daily and NA (either ETV 0.5 mg, TDF 300 mg, or TAF 25 mg) tablet orally once daily up to 48 weeks during double-blind phase. Participants who met NA treatment completion criteria at Week 48 that is ALT <3*ULN, HBV DNA < LLOQ, HBeAg negative, HBsAg <10 IU/mL entered follow up phase 1: participants who did not meet NA treatment completion criteria or did not stop NA, follow up phase 2: participants who Met NA treatment completion criteria at Week 44 and stopped NA at Week 48, follow up phase 3: participants who met NA treatment completion criteria after Week 44 and stopped NA during follow-up and were monitored closely for 48 weeks. Participants who did not meet above criteria at Week 48 continued NA treatment during 48-week follow-up phase. Participants who completed NA treatment during the follow-up phase entered the extended follow up phase up to 48 weeks (extended follow up Week 1 to extended follow up Week 48).
- Arm 4: JNJ-73763989 40 mg + Placebo + NA: Participants with CHB received JNJ-73763989 40 mg as SC injection once every 4 weeks along with placebo matching to JNJ-56136379 tablet orally once daily and NA (either ETV 0.5 mg, TDF 300 mg, or TAF 25 mg) tablet orally once daily up to 48 weeks during double blind phase. Participants who met NA treatment completion criteria at Week 48 that is ALT <3*ULN, HBV DNA < LLOQ, HBeAg negative, HBsAg <10 IU/mL entered follow up phase 1: participants who did not meet NA treatment completion criteria or did not stop NA, follow up phase 2: participants who Met NA treatment completion criteria at Week 44 and stopped NA at Week 48, follow up phase 3: participants who met NA treatment completion criteria after Week 44 and stopped NA during follow-up and were monitored closely for 48 weeks. Participants who did not meet above criteria at Week 48 continued NA treatment during 48-week follow-up phase. Participants who completed NA treatment during the follow-up phase entered the extended follow up phase up to 48 weeks (extended follow up Week 1 to extended follow up Week 48).
- Arm 5: Placebo + JNJ-56136379 250 mg + NA: Participants with CHB received placebo matching to JNJ-73763989 as SC injection once every 4 weeks and a fixed dose of JNJ-56136379 250 mg oral tablet once daily along with NA (either ETV 0.5 mg, TDF 300 mg, or TAF 25 mg) tablet orally once daily up to 48 weeks during double blind phase. Participants who met NA treatment completion criteria at Week 48 that is ALT <3*ULN, HBV DNA < LLOQ, HBeAg negative, HBsAg <10 IU/mL entered follow up phase 1: participants who did not meet NA treatment completion criteria or did not stop NA, follow up phase 2: participants who Met NA treatment completion criteria at Week 44 and stopped NA at Week 48, follow up phase 3: participants who met NA treatment completion criteria after Week 44 and stopped NA during follow-up and were monitored closely for 48 weeks. Participants who did not meet above criteria at Week 48 continued NA treatment during 48-week follow-up phase. Participants who completed NA treatment during the follow-up phase entered the extended follow up phase up to 48 weeks (extended follow up Week 1 to extended follow up Week 48).
- Arm 6: Placebo + Placebo + NA: Participants with CHB received placebo matching to JNJ-73763989 as SC injection once every 4 weeks and placebo matching to JNJ-56136379 tablet orally once daily along with NA (either ETV 0.5 mg, TDF 300 mg, or TAF 25 mg) tablet orally once daily up to 48 weeks during double blind phase. Participants who met NA treatment completion criteria at Week 48 that is ALT <3*ULN, HBV DNA < LLOQ, HBeAg negative, HBsAg <10 IU/mL entered follow up phase 1: participants who did not meet NA treatment completion criteria or did not stop NA, follow up phase 2: participants who Met NA treatment completion criteria at Week 44 and stopped NA at Week 48, follow up phase 3: participants who met NA treatment completion criteria after Week 44 and stopped NA during follow-up and were monitored closely for 48 weeks. Participants who did not meet above criteria at Week 48 continued NA treatment during 48-week follow-up phase. Participants who completed NA treatment during the follow-up phase entered the extended follow up phase up to 48 weeks (extended follow up Week 1 to extended follow up Week 48).
Period: Overall Study
Arm/Group | Arm 1: JNJ-73763989 100 mg + JNJ-56136379 250 mg + NA | Arm 2: JNJ-73763989 200 mg + Placebo + NA | Arm 3: JNJ-73763989 100 mg + Placebo + NA | Arm 4: JNJ-73763989 40 mg + Placebo + NA | Arm 5: Placebo + JNJ-56136379 250 mg + NA | Arm 6: Placebo + Placebo + NA
Started | 95 | 96 | 93 | 94 | 48 | 45
Double Blind Phase | 95 | 96 | 93 | 93 | 48 | 45
Follow up Phase 1: (Included participants who did not meet NA treatment completion criteria or did not stop NA) | 81 | 70 | 71 | 85 | 47 | 44
Follow up Phase 2: (Included participants who met NA treatment completion criteria at Week 44 and stopped NA at Week 48) | 8 | 17 | 15 | 5 | 0 | 1
Follow up Phase 3: (Included participants who met NA treatment completion criteria after Week 44 and stopped NA during follow-up) | 3 | 8 | 5 | 0 | 0 | 0
Extended Follow up (Included participants who completed NA treatment during the follow-up phase) | 3 | 7 | 5 | 0 | 0 | 0
Treated | 95 | 96 | 93 | 94 | 48 | 45
Completed | 92 | 90 | 90 | 85 | 45 | 45
Not Completed | 3 | 6 | 3 | 9 | 3 | 0
Not completed — Lost to Follow-up | 0 | 1 | 2 | 1 | 1 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 4 | 1 | 7 | 2 | 0
Not completed — Randomized and not treated | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intent to treat (ITT) set included all participants who were randomly assigned to any of the 6 intervention arms and received at least 1 dose of study intervention.
Groups:
- Arm 1: JNJ-73763989 (100 mg) + JNJ-56136379 (250 mg) + NA Participants Received: Participants with chronic hepatitis B (CHB) received JNJ-73763989 100 milligrams (mg) as subcutaneous (SC) injection once every 4 weeks along with JNJ-56136379 250 mg as oral tablet once daily and Nucleos(t)ide Analog (NA) (either entecavir [ETV] monohydrate 0.5 mg, tenofovir disoproxil fumarate [TDF] 300 mg, or tenofovir alafenamide [TAF] 25 mg) tablet orally once daily up to 48 weeks during double blind phase. Participants who met NA treatment completion criteria at Week 48 that is alanine aminotransferase (ALT) less than (<) 3*upper limit of normal (ULN), hepatitis B virus (HBV) deoxyribonucleic acid (DNA) < lower limit of quantification (LLOQ), hepatitis B e antigen (HBeAg) negative, hepatitis B surface antigen (HBsAg) less than (<) 10 international unit per milliliter (IU/mL) entered follow up phase 1: participants who did not meet NA treatment completion criteria or did not stop NA, follow up phase 2: participants who Met NA treatment completion criteria at Week 44 and stopped NA at Week 48, follow up phase 3: participants who met NA treatment completion criteria after Week 44 and stopped NA during follow-up and were monitored closely for 48 weeks. Participants who did not meet above criteria at Week 48 continued NA treatment during 48-week follow-up phase. Participants who completed NA treatment during the follow-up phase entered the extended follow up phase up to 48 weeks (extended follow up Week 1 to extended follow up Week 48).
- Total: Total of all reporting groups
Arm/Group | Arm 1: JNJ-73763989 (100 mg) + JNJ-56136379 (250 mg) + NA Participants Received | Arm 2: JNJ-73763989 200 mg + Placebo + NA | Arm 3: JNJ-73763989 100 mg + Placebo + NA | Arm 4: JNJ-73763989 40 mg + Placebo + NA | Arm 5: Placebo + JNJ-56136379 250 mg + NA | Arm 6: Placebo + Placebo + NA | Total
Number analyzed (Participants) | 95 | 96 | 93 | 93 | 48 | 45 | 470
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.8 (10.72) | 42.9 (10.9) | 43 (11.3) | 42.2 (10.92) | 43.9 (9.8) | 43.8 (9.99) | 43.0 (10.71)
Age, Customized [Count of Participants; unit: Participants]
  Children (2-11 years) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Adolescents (12-17 years) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Adults (18-64 years) | 94 | 95 | 89 | 93 | 46 | 45 | 462
  From 65 to 84 years | 1 | 1 | 4 | 0 | 2 | 0 | 8
  85 years and over | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 35 | 38 | 32 | 11 | 20 | 160
  Male | 71 | 61 | 55 | 61 | 37 | 25 | 310
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 2 | 1 | 0 | 3
  Asian | 35 | 39 | 39 | 42 | 20 | 15 | 190
  Black or African American | 6 | 7 | 5 | 9 | 2 | 1 | 30
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 54 | 50 | 48 | 39 | 25 | 28 | 244
  Unknown or not reported | 0 | 0 | 1 | 1 | 0 | 1 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  BELGIUM | 4 | 4 | 3 | 5 | 1 | 2 | 19
  BRAZIL | 1 | 2 | 0 | 1 | 0 | 0 | 4
  CANADA | 3 | 4 | 6 | 4 | 2 | 1 | 20
  CHINA | 1 | 0 | 4 | 1 | 0 | 0 | 6
  CZECH REPUBLIC | 9 | 8 | 2 | 3 | 3 | 2 | 27
  FRANCE | 4 | 7 | 3 | 4 | 4 | 0 | 22
  GERMANY | 6 | 5 | 2 | 1 | 2 | 0 | 16
  ITALY | 6 | 7 | 4 | 5 | 3 | 5 | 30
  JAPAN | 10 | 12 | 13 | 18 | 6 | 2 | 61
  MALAYSIA | 2 | 5 | 2 | 3 | 3 | 3 | 18
  POLAND | 8 | 8 | 8 | 6 | 2 | 5 | 37
  RUSSIAN FEDERATION | 12 | 8 | 13 | 13 | 11 | 5 | 62
  SOUTH KOREA | 2 | 2 | 0 | 3 | 1 | 2 | 10
  SPAIN | 5 | 1 | 5 | 8 | 0 | 3 | 22
  THAILAND | 6 | 5 | 5 | 4 | 2 | 1 | 23
  TURKEY | 11 | 10 | 12 | 6 | 3 | 7 | 49
  UNITED KINGDOM | 1 | 3 | 1 | 3 | 2 | 2 | 12
  UNITED STATES | 1 | 3 | 6 | 5 | 3 | 3 | 21
  Hong Kong, S.A.R., China | 3 | 2 | 4 | 0 | 0 | 2 | 11

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Meeting the Nucleos(t)Ide Analog (NA) Treatment Completion Criteria at Week 48
Description: Percentage of participants meeting the NA treatment completion criteria at Week 48 were reported. A participant was defined as a responder in meeting the NA treatment completion criteria at Week 48, if the following criteria were met based on the clinical laboratory tests performed at Week 44: participants had alanine transaminase (ALT) less than (<) 3*upper limit of normal range (ULN); had hepatitis B virus deoxyribonucleic acid (HBV DNA) < lower limit of quantification (LLOQ); was hepatitis B e antigen (HBeAg)-negative; had hepatitis B surface antigen (HBsAg) <10 international units per milliliter (IU/mL). Multiple Imputation using a longitudinal multiple regression model was applied to impute missing data.
Time Frame: Week 48
Population: Modified Intent-to-Treat (mITT) set was defined as all participants who were randomized in the study and received at least one dose of study treatment excluding those participants impacted by the COVID-19 pandemic defined as those participants who, because of COVID-19 or similar pandemic-related reasons, withdrew prematurely from the study prior to Week 44, or had no efficacy assessment for the primary outcome measure.
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm 1: JNJ-73763989 100 mg + JNJ-56136379 250 mg + NA | Arm 2: JNJ-73763989 200 mg + Placebo + NA | Arm 3: JNJ-73763989 100 mg + Placebo + NA | Arm 4: JNJ-73763989 40 mg + Placebo + NA | Arm 5: Placebo + JNJ-56136379 250 mg + NA | Arm 6: Placebo + Placebo + NA
Number analyzed (Participants) | 94 | 94 | 92 | 91 | 48 | 45
Percentage of participants | 9.4 (4.36) [4.36 to 14.36] | 19.1 (12.76) [12.76 to 27.06] | 16.3 (10.33) [10.33 to 23.99] | 5.5 (2.19) [2.19 to 11.21] | 0.0 (0.00) [0.00 to 6.05] | 2.2 (0.11) [0.11 to 10.11]
Statistical Analysis 1: Comparison: Arm 5: Placebo + JNJ-56136379 250 mg + NA vs Arm 6: Placebo + Placebo + NA; Test type: Superiority; p = 0.848, Mantel Haenszel; Difference of proportions = -2.3, 90% CI 2-sided [-5.97 to 1.38]
Statistical Analysis 2: Comparison: Arm 1: JNJ-73763989 100 mg + JNJ-56136379 250 mg + NA vs Arm 6: Placebo + Placebo + NA; Test type: Superiority; p = 0.027, Mantel Haenszel; Difference of proportions = 7.4, 90% CI 2-sided [1.07 to 13.68]
Statistical Analysis 3: Comparison: Arm 1: JNJ-73763989 100 mg + JNJ-56136379 250 mg + NA vs Arm 5: Placebo + JNJ-56136379 250 mg + NA; Test type: Superiority; p = 0.917, Mantel Haenszel; Difference of proportions = 9.1, 90% CI 2-sided [4.16 to 14.07]
Statistical Analysis 4: Comparison: Arm 1: JNJ-73763989 100 mg + JNJ-56136379 250 mg + NA vs Arm 3: JNJ-73763989 100 mg + Placebo + NA; Test type: Superiority; p = 0.917, Mantel Haenszel; Difference of proportions = -6.7, 90% CI 2-sided [-14.67 to 1.25]

2. Secondary Outcome: Double-blind Phase: Percentage of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An AE was any untoward medical occurrence in a clinical study participants administered a medicinal (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the intervention. Treatment-emergent AEs were defined as AEs with onset or worsening on or after date of first dose of study treatment.
Time Frame: Baseline up to Week 48
Population: Safety analysis set included all participants who received at least one dose of any of the study treatments.
Measure: Number; unit: Percentage of participants
Groups:
- Arm 1: DB Phase: JNJ-73763989 100 mg + JNJ-56136379 250 mg + NA: Participants with chronic hepatitis B (CHB) received JNJ-73763989 100 milligrams (mg) as subcutaneous (SC) injection once every 4 weeks along with JNJ-56136379 250 mg as oral tablet once daily and Nucleos(t)ide Analog (NA) (either entecavir [ETV] monohydrate 0.5 mg, tenofovir disoproxil fumarate [TDF] 300 mg, or tenofovir alafenamide [TAF] 25 mg) tablet orally once daily up to 48 weeks during double blind phase.
- Arm 2: DB Phase: JNJ-73763989 200 mg + Placebo + NA: Participants with CHB received JNJ-73763989 200 mg as SC injection once every 4 weeks along with placebo matching to JNJ-56136379 tablet orally once daily and NA (either ETV 0.5 mg, TDF 300 mg, or TAF 25 mg) tablet orally once daily up to 48 weeks during double blind phase.
- Arm 3: DB Phase: JNJ-73763989 100 mg + Placebo + NA: Participants with CHB received JNJ-73763989 100 mg as SC injection once every 4 weeks along with placebo matching to JNJ-56136379 tablet orally once daily and NA (either ETV 0.5 mg, TDF 300 mg, or TAF 25 mg) tablet orally once daily up to 48 weeks during double-blind phase.
- Arm 4: DB Phase: JNJ-73763989 40 mg + Placebo + NA: Participants with CHB received JNJ-73763989 40 mg as SC injection once every 4 weeks along with placebo matching to JNJ-56136379 tablet orally once daily and NA (either ETV 0.5 mg, TDF 300 mg, or TAF 25 mg) tablet orally once daily up to 48 weeks during double blind phase.
- Arm 5: DB Phase: Placebo + JNJ-56136379 250 mg + NA: Participants with CHB received placebo matching to JNJ-73763989 as SC injection once every 4 weeks and a fixed dose of JNJ-56136379 250 mg oral tablet once daily along with NA (either ETV 0.5 mg, TDF 300 mg, or TAF 25 mg) tablet orally once daily up to 48 weeks during double blind phase.
- Arm 6: DB Phase: Placebo + Placebo + NA: Participants with CHB received placebo matching to JNJ-73763989 as SC injection once every 4 weeks and placebo matching to JNJ-56136379 tablet orally once daily along with NA (either ETV 0.5 mg, TDF 300 mg, or TAF 25 mg) tablet orally once daily up to 48 weeks during double blind phase.
Arm/Group | Arm 1: DB Phase: JNJ-73763989 100 mg + JNJ-56136379 250 mg + NA | Arm 2: DB Phase: JNJ-73763989 200 mg + Placebo + NA | Arm 3: DB Phase: JNJ-73763989 100 mg + Placebo + NA | Arm 4: DB Phase: JNJ-73763989 40 mg + Placebo + NA | Arm 5: DB Phase: Placebo + JNJ-56136379 250 mg + NA | Arm 6: DB Phase: Placebo + Placebo + NA
Number analyzed (Participants) | 95 | 96 | 93 | 93 | 48 | 45
Percentage of participants | 71.6 | 64.6 | 71.0 | 74.2 | 85.4 | 66.7

3. Secondary Outcome: Follow-up Phase 1: Percentage of Participants With TEAEs
Description: as for outcome 2
Time Frame: From Week 48 up to Week 96
Population: Safety analysis set included all participants who received at least one dose of any of the study treatments.
Measure: Number; unit: Percentage of participants
Groups:
- Arm 1: Follow up Phase 1: JNJ-73763989 (100 mg) + JNJ-56136379 (250 mg) + NA: Participants who received JNJ-73763989 100 mg) as SC injection once every 4 weeks along with JNJ-56136379 250 mg as oral tablet once daily and NA (either ETV monohydrate 0.5 mg, TDF 300 mg, or TAF 25 mg) tablet orally once daily up to 48 weeks during double blind phase and did not meet NA treatment completion criteria or did not stop NA were followed-up till Week 96.
- Arm 2: Follow up Phase 1: JNJ-73763989 (200mg) + Placebo + NA: Participants who received JNJ-73763989 along with placebo matching to JNJ-56136379 and NA up to 48 weeks during double blind phase and did Not meet NA treatment completion criteria or did not stop NA were followed-up till Week 96.
- Arm 3: Follow up Phase 1: JNJ-73763989 (100 mg) + Placebo + NA: Participants who received JNJ-73763989 100 along with placebo matching to JNJ-56136379 and NA up to 48 weeks during double blind phase and and did Not meet NA treatment completion criteria or did not stop NA were followed-up till Week 96.
- Arm 4: Follow up Phase 1: JNJ-73763989 (40 mg) + Placebo + NA: Participants who received JNJ-73763989 40 mg along with placebo matching to JNJ-56136379 and NA up to 48 weeks in double blind phase and and did Not meet NA treatment completion criteria or did not stop NA were followed-up till Week 96.
- Arm 5: Follow up Phase 1: Placebo + JNJ-56136379 250 mg + NA: Participants who received placebo matching to JNJ-73763989 along with a fixed dose of JNJ-56136379 250 mg and NA up to 48 weeks during the double blind phase and did Not meet NA treatment completion criteria or did not stop NA were followed-up till Week 96.
- Arm 6 :Follow up Phase 1: Placebo + Placebo + NA: Participants who received placebo matching to JNJ-73763989 along with placebo matching to JNJ-56136379 and NA up to 48 weeks during the double blind phase and did not meet NA treatment completion criteria or did Not stop NA were followed up till week 96.
Arm/Group | Arm 1: Follow up Phase 1: JNJ-73763989 (100 mg) + JNJ-56136379 (250 mg) + NA | Arm 2: Follow up Phase 1: JNJ-73763989 (200mg) + Placebo + NA | Arm 3: Follow up Phase 1: JNJ-73763989 (100 mg) + Placebo + NA | Arm 4: Follow up Phase 1: JNJ-73763989 (40 mg) + Placebo + NA | Arm 5: Follow up Phase 1: Placebo + JNJ-56136379 250 mg + NA | Arm 6 :Follow up Phase 1: Placebo + Placebo + NA
Number analyzed (Participants) | 81 | 70 | 71 | 85 | 47 | 44
Percentage of participants | 48.1 | 45.7 | 56.3 | 44.7 | 55.3 | 31.8

4. Secondary Outcome: Follow-up Phase 2: Percentage of Participants With TEAEs
Description: as for outcome 2
Time Frame: From Week 48 up to Week 96
Population: Safety analysis set included all participants who received at least one dose of any of the study treatments. '0' in the number of participants analyzed field signifies that none of the participant from the double-blind phase entered the respective follow up phase.
Measure: Number; unit: Percentage of participants
Groups:
- Arm 1: Follow up Phase 2: JNJ-73763989 (100 mg) + JNJ-56136379 (250 mg) + NA: Participants who received JNJ-73763989 100 mg) along with JNJ-56136379 250 mg and NA up to 48 weeks during double blind period and who met NA treatment completion criteria at Week 44 and stopped NA at Week 48 were followed-up till Week 96.
- Arm 2: Follow up Phase 2: JNJ-73763989 (200mg) + Placebo + NA: Participants who received JNJ-73763989 100 mg along with JNJ-56136379 250 mg and NA up to 48 weeks during double blind period who met NA treatment completion criteria at Week 44 and stopped NA at Week 48 were followed-up till Week 96.
- Arm 3: Follow up Phase 2: JNJ-73763989 (100 mg) + Placebo + NA: Participants who received JNJ-73763989 100 along with placebo matching to JNJ-56136379 and NA up to 48 weeks during double blind phase and who met NA treatment completion criteria at Week 44 and stopped NA at Week 48 were followed-up till Week 96.
- Arm 4: Follow up Phase 2: JNJ-73763989 (40 mg) + Placebo + NA: Participants who received JNJ-73763989 along with placebo matching to JNJ-56136379 and NA up to 48 weeks during double blind phase and who met NA treatment completion criteria at Week 44 and stopped NA at Week 48 were followed-up till Week 96.
- Arm 5: Follow up Phase 2: Placebo + JNJ-56136379 250 mg + NA: Participants who received placebo matching to JNJ-73763989 along with a fixed dose of JNJ-56136379 250 mg and NA up to 48 weeks during the double blind phase and who met NA treatment completion criteria at Week 44 and stopped NA at Week 48 were followed-up till Week 96.
- Arm 6: Follow up Phase 2: Placebo + Placebo + NA: Participants who received placebo matching to JNJ-73763989 and placebo matching to JNJ-56136379 along with NA up to 48 weeks during double blind phase and who met NA treatment completion criteria at Week 44 and stopped NA at Week 48 were followed-up till Week 96.
Arm/Group | Arm 1: Follow up Phase 2: JNJ-73763989 (100 mg) + JNJ-56136379 (250 mg) + NA | Arm 2: Follow up Phase 2: JNJ-73763989 (200mg) + Placebo + NA | Arm 3: Follow up Phase 2: JNJ-73763989 (100 mg) + Placebo + NA | Arm 4: Follow up Phase 2: JNJ-73763989 (40 mg) + Placebo + NA | Arm 5: Follow up Phase 2: Placebo + JNJ-56136379 250 mg + NA | Arm 6: Follow up Phase 2: Placebo + Placebo + NA
Number analyzed (Participants) | 8 | 17 | 15 | 5 | 0 | 1
Percentage of participants | 37.5 | 29.4 | 60.0 | 60.0 |  | 0

5. Secondary Outcome: Follow-up Phase 3: Percentage of Participants With TEAEs
Description: as for outcome 2
Time Frame: From Week 48 up to Week 96
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Groups:
- Arm 1: Follow up Phase 3: JNJ-73763989 (100 mg) + JNJ-56136379 (250 mg) + NA: Participants who received JNJ-73763989 100 mg) as SC injection once every 4 weeks along with JNJ-56136379 250 mg as oral tablet once daily and NA (either ETV monohydrate 0.5 mg, TDF 300 mg, or TAF 25 mg) tablet orally once daily up to 48 weeks during the double blind phase and who met NA treatment completion criteria after Week 44 and stopped NA during Follow-up followed-up till Week 96.
- Arm 2: Follow up Period 3: JNJ-73763989 (200mg) + Placebo + NA: Participants received JNJ-73763989 200 mg along with placebo matching to JNJ-56136379 up to 48 weeks during double blind phase and who met NA treatment completion criteria after Week 44 and stopped NA during Follow-up were followed-up till Week 96.
- Arm 3: Follow up Phase 3: JNJ-73763989 (100 mg) + Placebo + NA: Participants received JNJ-73763989 100 mg along with placebo matching to JNJ-56136379 to 48 weeks during double blind phase and who met NA treatment completion criteria after Week 44 and Stopped NA during Follow-up followed-up till Week 96.
- Arm 4: Follow up Phase 3: JNJ-73763989 (40 mg) + Placebo + NA: Participants who received JNJ-73763989 40 mg along with placebo matching to JNJ-56136379 and NA up to 48 weeks during double blind phase and who met NA treatment completion criteria after Week 44 and Stopped NA during Follow-up were followed-up till Week 96.
- Arm 5: Follow up Phase 3: Placebo + JNJ-56136379 250 mg + NA: Participants who received placebo matching to JNJ-73763989 along with a fixed dose of JNJ-56136379 250 mg and NA up to 48 weeks during the double blind phase and who met NA treatment completion criteria after Week 44 and Stopped NA during Follow-up followed-up till Week 96.
- Arm 6: Follow up Phase 3: Placebo + Placebo + NA: Participants who received placebo matching to JNJ-73763989 along with placebo matching to JNJ-56136379 and NA up to 48 weeks during the double blind phase and who met NA treatment completion criteria after Week 44 and Stopped NA during Follow-up followed-up till Week 96.
Arm/Group | Arm 1: Follow up Phase 3: JNJ-73763989 (100 mg) + JNJ-56136379 (250 mg) + NA | Arm 2: Follow up Period 3: JNJ-73763989 (200mg) + Placebo + NA | Arm 3: Follow up Phase 3: JNJ-73763989 (100 mg) + Placebo + NA | Arm 4: Follow up Phase 3: JNJ-73763989 (40 mg) + Placebo + NA | Arm 5: Follow up Phase 3: Placebo + JNJ-56136379 250 mg + NA | Arm 6: Follow up Phase 3: Placebo + Placebo + NA
Number analyzed (Participants) | 3 | 8 | 5 | 0 | 0 | 0
Percentage of participants | 33.3 | 37.5 | 20.0 |  |  |

6. Secondary Outcome: Extended Follow-up Phase: Percentage of Participants With TEAEs
Description: as for outcome 2
Time Frame: Extended Follow up Week 1 to extended follow up Week 48
Population: Safety analysis set included all participants who received at least one dose of any of the study treatments. '0' in the number of participants analyzed field signifies that none of the participant from the follow up phase entered the extended follow up phase.
Measure: Number; unit: Percentage of participants
Groups:
- Arm 1: Extended Follow up: JNJ-73763989 (100 mg) + JNJ-56136379 (250 mg) + NA: Participants received JNJ-73763989 100 mg along with JNJ-56136379 250 mg NA up to 48 weeks during double blind phase. Participants who completed NA treatment during the follow-up phase and completed the assessments of the end of study visit were followed up for extended follow up Week 1 to extended follow up Week 48.
- Arm 2: Extended Follow Up: JNJ-73763989 (200 mg) + Placebo + NA: Participants received JNJ-73763989 200 mg along with placebo matching to JNJ-56136379 and NA up to 48 weeks during double blind phase. Participants who completed NA treatment during the follow-up phase and completed the assessments of the end of study visit were followed up for extended follow up Week 1 to extended follow up Week 48.
- Arm 3: Extended Follow up: JNJ-73763989 (100 mg) + Placebo + NA: Participants received JNJ-73763989 100 mg along with placebo matching to JNJ-56136379 NA up to 48 weeks during double blind phase. Participants who completed NA treatment during the follow-up phase and completed the assessments of the end of study visit were followed up for extended follow up Week 1 to extended follow up Week 48.
- Arm 4: Extended Follow Up: JNJ-73763989 (40 mg) + Placebo + NA: Participants received JNJ-73763989 40 mg along with placebo matching to JNJ-56136379 and NA up to 48 weeks in double blind phase. Participants who completed NA treatment during the follow-up phase and completed the assessments of the end of study visit were followed up for extended follow up Week 1 to extended follow up Week 48.
- Arm 5: Extended Follow Up: Placebo + JNJ-56136379 250 mg + NA: Participants received placebo matching to JNJ-73763989 along with a fixed dose of JNJ-56136379 250 mg and NA up to 48 weeks during the double blind phase. Participants who completed NA treatment during the follow-up phase and completed the assessments of the end of study visit were followed up for extended follow up Week 1 to extended follow up Week 48.
- Arm 6: Extended Follow Up: Placebo + Placebo + NA: Participants received placebo matching to JNJ-73763989 along with placebo matching to JNJ-56136379 and NA up to 48 weeks during the double blind phase. Participants who completed NA treatment during the follow-up phase and completed the assessments of the end of study visit were followed up for extended follow up Week 1 to extended follow up Week 48.
Arm/Group | Arm 1: Extended Follow up: JNJ-73763989 (100 mg) + JNJ-56136379 (250 mg) + NA | Arm 2: Extended Follow Up: JNJ-73763989 (200 mg) + Placebo + NA | Arm 3: Extended Follow up: JNJ-73763989 (100 mg) + Placebo + NA | Arm 4: Extended Follow Up: JNJ-73763989 (40 mg) + Placebo + NA | Arm 5: Extended Follow Up: Placebo + JNJ-56136379 250 mg + NA | Arm 6: Extended Follow Up: Placebo + Placebo + NA
Number analyzed (Participants) | 3 | 7 | 5 | 0 | 0 | 0
Percentage of participants | 66.7 | 71.4 | 100.0 |  |  |

7. Secondary Outcome: Double-blind Phase: Percentage of Participants With Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE was any untoward medical occurrence that at any dose may result in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, was a suspected transmission of any infectious agent via a medicinal product, and was medically important.
Time Frame: Baseline up to Week 48
Population: Safety analysis set included all participants who received at least one dose of any of the study treatments.
Measure: Number; unit: Percentage of participants
Arm/Group | Arm 1: DB Phase: JNJ-73763989 100 mg + JNJ-56136379 250 mg + NA | Arm 2: DB Phase: JNJ-73763989 200 mg + Placebo + NA | Arm 3: DB Phase: JNJ-73763989 100 mg + Placebo + NA | Arm 4: DB Phase: JNJ-73763989 40 mg + Placebo + NA | Arm 5: DB Phase: Placebo + JNJ-56136379 250 mg + NA | Arm 6: DB Phase: Placebo + Placebo + NA
Number analyzed (Participants) | 95 | 96 | 93 | 93 | 48 | 45
Percentage of participants | 2.1 | 3.1 | 2.2 | 1.1 | 4.2 | 0

8. Secondary Outcome: Follow-up Phase 1: Percentage of Participants With SAEs
Description: as for outcome 7
Time Frame: From Week 48 up to Week 96
Population: Safety analysis set included all participants who received at least one dose of any of the study treatments.
Measure: Number; unit: Percentage of participants
Groups:
- Arm 3: Follow up Phase 1: JNJ-73763989 (100 mg) + Placebo + NA: Participants who received JNJ-73763989 100 along with placebo matching to JNJ-56136379 and NA up to 48 weeks during double blind phase and Did Not meet NA treatment completion criteria or did not stop NA were followed-up till Week 96.
- Arm 4: Follow up Phase 1: JNJ-73763989 (40 mg) + Placebo + NA: Participants who received JNJ-73763989 40 mg along with placebo matching to JNJ-56136379 and NA up to 48 weeks in double blind phase and Did Not meet NA treatment completion criteria or did not stop NA were followed-up till Week 96.
- Arm 5: Follow up Phase 1: Placebo + JNJ-56136379 250 mg + NA: Participants who received placebo matching to JNJ-73763989 along with a fixed dose of JNJ-56136379 250 mg and NA up to 48 weeks during the double blind phase and Did Not meet NA treatment completion criteria or did not stop NA were followed-up tll Week 96.
Arm/Group | Arm 1: Follow up Phase 1: JNJ-73763989 (100 mg) + JNJ-56136379 (250 mg) + NA | Arm 2: Follow up Phase 1: JNJ-73763989 (200mg) + Placebo + NA | Arm 3: Follow up Phase 1: JNJ-73763989 (100 mg) + Placebo + NA | Arm 4: Follow up Phase 1: JNJ-73763989 (40 mg) + Placebo + NA | Arm 5: Follow up Phase 1: Placebo + JNJ-56136379 250 mg + NA | Arm 6 :Follow up Phase 1: Placebo + Placebo + NA
Number analyzed (Participants) | 81 | 70 | 71 | 85 | 47 | 44
Percentage of participants | 1.2 | 7.1 | 4.2 | 1.2 | 2.1 | 0

9. Secondary Outcome: Follow-up Phase 2: Percentage of Participants With SAEs
Description: as for outcome 7
Time Frame: From Week 48 up to Week 96
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Groups:
- Arm 2: Follow up Phase 2: JNJ-73763989 (200mg) + Placebo + NA: Participants who received JNJ-73763989 100 mg along with JNJ-56136379 250 mg and NA up to 48 weeks during double blind period and who met NA treatment completion criteria at Week 44 and stopped NA at Week 48 were followed-up till Week 96.
- Arm 3: Follow up Phase 2: JNJ-73763989 (100 mg) + Placebo + NA: Participants who received JNJ-73763989 100 along with placebo matching to JNJ-56136379 and NA up to 48 weeks during double blind phase and who met NA treatment completion criteria and stopped NA at Week 48 were followed-up till Week 96.
- Arm 4: Follow up Phase 2: JNJ-73763989 (40 mg) + Placebo + NA: Participants who received JNJ-73763989 along with placebo matching to JNJ-56136379 and NA up to 48 weeks during double blind phase and who met NA treatment completion criteria and stopped NA at Week 48 were followed-up till Week 96.
- Arm 5: Follow up Phase 2: Placebo + JNJ-56136379 250 mg + NA: Participants who received placebo matching to JNJ-73763989 along with a fixed dose of JNJ-56136379 250 mg and NA up to 48 weeks during the double blind phase and who met NA treatment completion criteria and stopped NA at Week 48 were followed-up till Week 96.
- Arm 6: Follow up Phase 2: Placebo + Placebo + NA: Participants who received placebo matching to JNJ-73763989 and placebo matching to JNJ-56136379 along with NA up to 48 weeks during double blind phase and who met NA treatment completion criteria and stopped NA at Week 48 were followed-up till Week 96.
Arm/Group | Arm 1: Follow up Phase 2: JNJ-73763989 (100 mg) + JNJ-56136379 (250 mg) + NA | Arm 2: Follow up Phase 2: JNJ-73763989 (200mg) + Placebo + NA | Arm 3: Follow up Phase 2: JNJ-73763989 (100 mg) + Placebo + NA | Arm 4: Follow up Phase 2: JNJ-73763989 (40 mg) + Placebo + NA | Arm 5: Follow up Phase 2: Placebo + JNJ-56136379 250 mg + NA | Arm 6: Follow up Phase 2: Placebo + Placebo + NA
Number analyzed (Participants) | 8 | 17 | 15 | 5 | 0 | 1
Percentage of participants | 12.5 | 0 | 0 | 0 |  | 0

10. Secondary Outcome: Follow-up Phase 3: Percentage of Participants With SAEs
Description: as for outcome 7
Time Frame: From Week 48 up to Week 96
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Groups:
- Arm 1: Follow up Phase 3: JNJ-73763989 (100 mg) + JNJ-56136379 (250 mg) + NA: Participants who received JNJ-73763989 100 mg) as SC injection once every 4 weeks along with JNJ-56136379 250 mg as oral tablet once daily and NA (either ETV monohydrate 0.5 mg, TDF 300 mg, or TAF 25 mg) tablet orally once daily up to 48 weeks and who met NA treatment completion criteria after Week 44 and Stopped NA during Follow-up followed-up till Week 96.
- Arm 4: Follow up Phase 3: JNJ-73763989 (40 mg) + Placebo + NA: Participants who received JNJ-73763989 40 mg along with placebo matching to JNJ-56136379 and NA up to 48 weeks in double blind phase and who met NA treatment completion criteria after Week 44 and Stopped NA during Follow-up were followed-up till Week 96.
Arm/Group | Arm 1: Follow up Phase 3: JNJ-73763989 (100 mg) + JNJ-56136379 (250 mg) + NA | Arm 2: Follow up Period 3: JNJ-73763989 (200mg) + Placebo + NA | Arm 3: Follow up Phase 3: JNJ-73763989 (100 mg) + Placebo + NA | Arm 4: Follow up Phase 3: JNJ-73763989 (40 mg) + Placebo + NA | Arm 5: Follow up Phase 3: Placebo + JNJ-56136379 250 mg + NA | Arm 6: Follow up Phase 3: Placebo + Placebo + NA
Number analyzed (Participants) | 3 | 8 | 5 | 0 | 0 | 0
Percentage of participants | 33.3 | 0 | 0 |  |  |

11. Secondary Outcome: Extended Follow-up Phase: Percentage of Participants With SAEs
Description: as for outcome 7
Time Frame: Extended Follow up Week 1 to extended follow up Week 48
Population: as for outcome 6
Measure: Number; unit: Percentage of participants
Groups:
- Arm 2: Extended Follow Up: JNJ-73763989 (200mg) + Placebo + NA: Participants received JNJ-73763989 200 mg along with placebo matching to JNJ-56136379 and NA up to 48 weeks during double blind phase. Participants who completed NA treatment during the follow-up phase and completed the assessments of the end of study visit were followed up for extended follow up Week 1 to extended follow up Week 48.
Arm/Group | Arm 1: Extended Follow up: JNJ-73763989 (100 mg) + JNJ-56136379 (250 mg) + NA | Arm 2: Extended Follow Up: JNJ-73763989 (200mg) + Placebo + NA | Arm 3: Extended Follow up: JNJ-73763989 (100 mg) + Placebo + NA | Arm 4: Extended Follow Up: JNJ-73763989 (40 mg) + Placebo + NA | Arm 5: Extended Follow Up: Placebo + JNJ-56136379 250 mg + NA | Arm 6: Extended Follow Up: Placebo + Placebo + NA
Number analyzed (Participants) | 3 | 7 | 5 | 0 | 0 | 0
Percentage of participants | 0 | 14.3 | 40.0 |  |  |

12. Secondary Outcome: Percentage of Participants With Abnormalities in Clinical Laboratory Tests (Hematology)
Description: Percentage of participants with abnormalities in clinical laboratory tests (hematology: Abnormally low [AL] and Abnormally high [AH] basophils, eosinophils, erthrocytes mean corpuscular hemoglobin concentration, erthrocytes mean corpuscular heamoglobin, erthrocytes mean corpuscular volume, erthrocytes, hematocrit, lymphocytes atypical, metamyelocytes, monocytes, myelocytes, neutrophils, segmented, reticulocytes) were reported. Abnormality was determined at the investigator's discretion. Here, M.C: Mean corpuscular. Participants with abnormally low or high values were reported.
Time Frame: Double blind (DB) phase: Baseline (Day 1) up to Week 48, Follow up (FU) phase: Week 48 up to Week 96
Population: Safety analysis set included all participants who received at least one dose of any of study treatments. Here, 'n' (number analyzed) represents number of participants evaluable at specified categories. Here 'n=0' signifies no participants were available for analysis at specified timepoints.
Measure: Number; unit: Percentage of participants
Arm/Group | Arm 1: JNJ-73763989 100 mg + JNJ-56136379 250 mg + NA | Arm 2: JNJ-73763989 200 mg + Placebo + NA | Arm 3: JNJ-73763989 100 mg + Placebo + NA | Arm 4: JNJ-73763989 40 mg + Placebo + NA | Arm 5: Placebo + JNJ-56136379 250 mg + NA | Arm 6: Placebo + Placebo + NA
Number analyzed (Participants) | 93 | 94 | 93 | 92 | 48 | 45
Percentage of participants
  DB:Basophils AL | 0 | 0 | 0 | 0 | 0 | 0
  DB:Basophils AH | 1.1 | 2.1 | 1.1 | 2.2 | 2.1 | 0
  F-U:Basophils AL: number analyzed (Participants) | 93 | 92 | 90 | 87 | 46 | 44
  F-U:Basophils AL | 0 | 0 | 0 | 0 | 0 | 0
  F-U:Basophils AH: number analyzed (Participants) | 93 | 92 | 90 | 87 | 46 | 44
  F-U:Basophils AH | 2.2 | 0 | 1.1 | 0 | 0 | 0
  DB:Eosinophils AL | 0 | 0 | 0 | 0 | 0 | 0
  DB:Eosinophils AH | 3.2 | 0 | 1.1 | 3.3 | 14.6 | 2.2
  F-U:Eosinophils AL: number analyzed (Participants) | 93 | 92 | 90 | 87 | 46 | 44
  F-U:Eosinophils AL | 0 | 0 | 0 | 0 | 0 | 0
  F-U:Eosinophils AH: number analyzed (Participants) | 93 | 92 | 90 | 87 | 46 | 44
  F-U:Eosinophils AH | 1.1 | 1.1 | 1.1 | 1.1 | 2.2 | 0
  DB:Ery. M.C HGB Conc. AL | 10.8 | 13.8 | 26.9 | 14.1 | 16.7 | 22.2
  DB:Ery. M.C HGB Conc. AH | 0 | 0 | 0 | 0 | 0 | 0
  F-U:Ery. M.C HGB Conc. AL: number analyzed (Participants) | 93 | 92 | 90 | 87 | 46 | 44
  F-U:Ery. M.C HGB Conc. AL | 13.0 | 17.4 | 24.4 | 18.4 | 13.0 | 22.7
  F-U:Ery. M.C HGB Conc. AH: number analyzed (Participants) | 93 | 92 | 90 | 87 | 46 | 44
  F-U:Ery. M.C HGB Conc. AH | 0 | 0 | 0 | 0 | 0 | 0
  DB:Ery. M.C Hemoglobin AL | 3.2 | 4.3 | 7.5 | 6.5 | 6.3 | 11.1
  DB:Ery. M.C Hemoglobin AH | 7.5 | 1.1 | 1.1 | 1.1 | 6.3 | 2.2
  F-U::Ery. M.C Hemoglobin AL: number analyzed (Participants) | 93 | 92 | 90 | 87 | 46 | 44
  F-U::Ery. M.C Hemoglobin AL | 7.5 | 8.7 | 6.7 | 8.0 | 2.2 | 6.8
  F-U::Ery. M.C Hemoglobin AH: number analyzed (Participants) | 93 | 92 | 90 | 87 | 46 | 44
  F-U::Ery. M.C Hemoglobin AH | 4.3 | 1.1 | 0 | 1.1 | 2.2 | 2.3
  DB:Ery. M.C Volume AL | 3.2 | 4.3 | 7.5 | 6.5 | 6.3 | 8.9
  DB:Ery. M.C Volume AH | 29.0 | 19.1 | 15.1 | 16.3 | 29.2 | 13.3
  F-U:Ery. M.C Volume AL: number analyzed (Participants) | 93 | 92 | 90 | 87 | 46 | 44
  F-U:Ery. M.C Volume AL | 4.3 | 6.5 | 7.8 | 6.9 | 2.2 | 4.5
  F-U:Ery. M.C Volume AH: number analyzed (Participants) | 93 | 92 | 90 | 87 | 46 | 44
  F-U:Ery. M.C Volume AH | 16.3 | 12.0 | 13.3 | 13.8 | 19.6 | 9.1
  DB:Erythrocytes AL | 20.4 | 14.9 | 24.7 | 15.2 | 27.1 | 22.2
  DB:Erythrocytes AH | 0 | 0 | 3.2 | 3.3 | 0 | 2.2
  F-U:Erythrocytes AL: number analyzed (Participants) | 93 | 92 | 90 | 87 | 46 | 44
  F-U:Erythrocytes AL | 18.3 | 13.0 | 21.1 | 19.5 | 21.7 | 13.6
  F-U:Erythrocytes AH: number analyzed (Participants) | 93 | 92 | 90 | 87 | 46 | 44
  F-U:Erythrocytes AH | 0 | 0 | 1.1 | 3.4 | 0 | 0
  DB:Hematocrit AL | 7.5 | 10.6 | 14.0 | 8.7 | 10.4 | 13.3
  DB:Hematocrit AH | 1.1 | 0 | 1.1 | 0 | 2.1 | 2.2
  F-U:Hematocrit AL: number analyzed (Participants) | 93 | 92 | 90 | 87 | 46 | 44
  F-U:Hematocrit AL | 6.5 | 13.0 | 10.0 | 11.5 | 13.0 | 11.4
  F-U: Hematocrit AH: number analyzed (Participants) | 93 | 92 | 90 | 87 | 46 | 44
  F-U: Hematocrit AH | 1.1 | 1.1 | 0 | 0 | 0 | 0
  DB:Lymphocytes Atypical AL: number analyzed (Participants) | 5 | 6 | 2 | 4 | 2 | 2
  DB:Lymphocytes Atypical AL | 0 | 0 | 0 | 0 | 0 | 0
  DB:Lymphocytes Atypical AH: number analyzed (Participants) | 5 | 6 | 2 | 4 | 2 | 2
  DB:Lymphocytes Atypical AH | 80.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0
  F-U:Lymphocytes Atypical AL: number analyzed (Participants) | 2 | 4 | 1 | 0 | 2 | 0
  F-U:Lymphocytes Atypical AL | 0 | 0 | 0 |  | 0 |
  F-U:Lymphocytes Atypical AH: number analyzed (Participants) | 2 | 4 | 1 | 0 | 2 | 0
  F-U:Lymphocytes Atypical AH | 100.0 | 100.0 | 100.0 |  | 100.0 |
  DB:Lymphocyte Atypical/Leukocyte AL: number analyzed (Participants) | 5 | 6 | 2 | 4 | 2 | 1
  DB:Lymphocyte Atypical/Leukocyte AL | 0 | 0 | 0 | 0 | 0 | 0
  DB:Lymphocyte Atypical/Leukocyte AH: number analyzed (Participants) | 5 | 6 | 2 | 4 | 2 | 1
  DB:Lymphocyte Atypical/Leukocyte AH | 80.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0
  F-U:LymphocyteAtypical/Leukocyte AL: number analyzed (Participants) | 2 | 4 | 1 | 0 | 1 | 0
  F-U:LymphocyteAtypical/Leukocyte AL | 0 | 0 | 0 |  | 0 |
  F-U:LymphocyteAtypical/Leukocyte AH: number analyzed (Participants) | 2 | 4 | 1 | 0 | 1 | 0
  F-U:LymphocyteAtypical/Leukocyte AH | 100.0 | 100.0 | 100.0 |  | 100.0 |
  F-U:Metamyelocytes AL: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0
  F-U:Metamyelocytes AL | 0 |  |  |  |  |
  F-U:Metamyelocytes AH: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0
  F-U:Metamyelocytes AH | 100.0 |  |  |  |  |
  DB:Monocytes AL | 10.8 | 12.8 | 5.4 | 5.4 | 4.2 | 8.9
  DB:Monocytes AH | 1.1 | 2.1 | 0 | 0 | 6.3 | 0
  F-U:Monocytes AL: number analyzed (Participants) | 93 | 92 | 90 | 87 | 46 | 44
  F-U:Monocytes AL | 4.3 | 7.6 | 7.8 | 1.1 | 4.3 | 0
  F-U:Monocytes AH: number analyzed (Participants) | 93 | 92 | 90 | 87 | 46 | 44
  F-U:Monocytes AH | 0 | 1.1 | 1.1 | 0 | 0 | 0
  F-U:Myelocytes AL: number analyzed (Participants) | 1 | 0 | 1 | 0 | 0 | 0
  F-U:Myelocytes AL | 0 |  | 0 |  |  |
  F-U:Myelocytes AH: number analyzed (Participants) | 1 | 0 | 1 | 0 | 0 | 0
  F-U:Myelocytes AH | 100.0 |  | 100.0 |  |  |
  DB:Neutrophils, Segmented AL | 36.6 | 24.5 | 23.7 | 25.0 | 35.4 | 33.3
  DB:Neutrophils, Segmented AH | 5.4 | 4.3 | 6.5 | 6.5 | 4.2 | 4.4
  F-U:Neutrophils,Segmented AL: number analyzed (Participants) | 93 | 92 | 90 | 87 | 46 | 44
  F-U:Neutrophils,Segmented AL | 30.1 | 23.9 | 18.9 | 26.4 | 17.4 | 20.5
  F-U:Neutrophils,Segmented AH: number analyzed (Participants) | 93 | 92 | 90 | 87 | 46 | 44
  F-U:Neutrophils,Segmented AH | 3.2 | 4.3 | 2.2 | 2.3 | 4.3 | 0
  DB:Reticulocytes AL: number analyzed (Participants) | 91 | 92 | 91 | 89 | 46 | 45
  DB:Reticulocytes AL | 34.1 | 27.2 | 26.4 | 24.7 | 41.3 | 37.8
  DB:Reticulocytes AH: number analyzed (Participants) | 91 | 92 | 91 | 89 | 46 | 45
  DB:Reticulocytes AH | 4.4 | 0 | 0 | 2.2 | 0 | 2.2
  F-U:Reticulocytes AL: number analyzed (Participants) | 92 | 92 | 90 | 86 | 46 | 44
  F-U:Reticulocytes AL | 27.2 | 32.6 | 24.4 | 20.9 | 30.4 | 13.6
  F-U:Reticulocytes AH: number analyzed (Participants) | 92 | 92 | 90 | 86 | 46 | 44
  F-U:Reticulocytes AH | 3.3 | 4.3 | 4.4 | 1.2 | 0 | 2.3

13. Secondary Outcome: Percentage of Participants With Abnormalities in Clinical Laboratory Tests (Chemistry)
Description: Percentage of participants with abnormalities in clinical laboratory tests (Chemistry: abnormally high and serum alpha fetoprotein, serum chloride, Serum gamma glutamyl tranferase [GGT], Serum high density cholesterol [HDL] Cholesterol, Indirect Bilirubin, Lactate Dehydrogenase, Serum Protein, Urea Nitrogen) were reported. Abnormality was determined at the investigator's discretion. Participants with abnormally low or high values were reported.
Time Frame: Double blind (DB) phase: Baseline up to Week 48, Follow up (FU) phase: Week 48 up to Week 96
Population: Safety analysis set included all participants who received at least one dose of any of study treatments. Here, 'n' (number analyzed) represents number of participants evaluable at specified categories and "N" (number of participants analyzed) represents number of participants evaluable for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Arm 1: JNJ-73763989 100 mg + JNJ-56136379 250 mg + NA | Arm 2: JNJ-73763989 200 mg + Placebo + NA | Arm 3: JNJ-73763989 100 mg + Placebo + NA | Arm 4: JNJ-73763989 40 mg + Placebo + NA | Arm 5: Placebo + JNJ-56136379 250 mg + NA | Arm 6: Placebo + Placebo + NA
Number analyzed (Participants) | 94 | 96 | 93 | 93 | 48 | 45
Percentage of participants
  DB:Serum Alpha Fetoprotein AL: number analyzed (Participants) | 87 | 91 | 88 | 89 | 46 | 43
  DB:Serum Alpha Fetoprotein AL | 0 | 0 | 0 | 0 | 0 | 0
  DB:Serum Alpha Fetoprotein AH: number analyzed (Participants) | 87 | 91 | 88 | 89 | 46 | 43
  DB:Serum Alpha Fetoprotein AH | 1.1 | 3.3 | 0 | 0 | 0 | 0
  F-U:Serum AlphaFetoprotein AL: number analyzed (Participants) | 89 | 85 | 85 | 86 | 46 | 45
  F-U:Serum AlphaFetoprotein AL | 0 | 0 | 0 | 0 | 0 | 0
  F-U:Serum AlphaFetoprotein AH: number analyzed (Participants) | 89 | 85 | 85 | 86 | 46 | 45
  F-U:Serum AlphaFetoprotein AH | 1.1 | 2.4 | 0 | 1.2 | 0 | 0
  F-U:Serum Chloride AL: number analyzed (Participants) | 94 | 94 | 90 | 88 | 46 | 45
  F-U:Serum Chloride AL | 0 | 0 | 0 | 0 | 0 | 0
  F-U:Serum Chloride AH: number analyzed (Participants) | 94 | 94 | 90 | 88 | 46 | 45
  F-U:Serum Chloride AH | 1.1 | 2.1 | 1.1 | 0 | 0 | 0
  DB:Serum GGT AL: number analyzed (Participants) | 93 | 96 | 93 | 93 | 48 | 45
  DB:Serum GGT AL | 1.1 | 3.1 | 5.4 | 8.6 | 2.1 | 8.9
  DB:Serum GGT AH: number analyzed (Participants) | 93 | 96 | 93 | 93 | 48 | 45
  DB:Serum GGT AH | 10.8 | 3.1 | 3.2 | 2.2 | 6.3 | 4.4
  F-U:Serum GGT AL: number analyzed (Participants) | 94 | 94 | 90 | 88 | 46 | 45
  F-U:Serum GGT AL | 1.1 | 3.2 | 3.3 | 9.1 | 8.7 | 4.4
  F-U:Serum GGT AH: number analyzed (Participants) | 94 | 94 | 90 | 88 | 46 | 45
  F-U:Serum GGT AH | 4.3 | 2.1 | 6.7 | 3.4 | 4.3 | 0
  DB:Serum HDL Cholesterol AL: number analyzed (Participants) | 93 | 96 | 93 | 93 | 48 | 45
  DB:Serum HDL Cholesterol AL | 6.5 | 18.8 | 24.7 | 28.0 | 8.3 | 37.8
  DB:Serum HDL Cholesterol AH: number analyzed (Participants) | 93 | 96 | 93 | 93 | 48 | 45
  DB:Serum HDL Cholesterol AH | 50.5 | 15.6 | 11.8 | 6.5 | 41.7 | 8.9
  F-U:Serum HDL Cholesterol AL: number analyzed (Participants) | 94 | 94 | 90 | 88 | 46 | 45
  F-U:Serum HDL Cholesterol AL | 18.1 | 20.2 | 15.6 | 28.4 | 19.6 | 17.8
  F-U:Serum HDL Cholesterol AH: number analyzed (Participants) | 94 | 94 | 90 | 88 | 46 | 45
  F-U:Serum HDL Cholesterol AH | 23.4 | 12.8 | 10.0 | 8.0 | 19.6 | 2.2
  DB:Indirect Bilirubin AL: number analyzed (Participants) | 93 | 96 | 93 | 93 | 48 | 45
  DB:Indirect Bilirubin AL | 0 | 0 | 0 | 0 | 0 | 0
  DB:Indirect Bilirubin AH: number analyzed (Participants) | 93 | 96 | 93 | 93 | 48 | 45
  DB:Indirect Bilirubin AH | 7.5 | 3.1 | 4.3 | 6.5 | 8.3 | 2.2
  F-U:Indirect Bilirubin AL: number analyzed (Participants) | 92 | 94 | 90 | 88 | 46 | 45
  F-U:Indirect Bilirubin AL | 0 | 0 | 0 | 0 | 0 | 0
  F-U:Indirect Bilirubin AH: number analyzed (Participants) | 92 | 94 | 90 | 88 | 46 | 45
  F-U:Indirect Bilirubin AH | 6.5 | 1.1 | 2.2 | 8.0 | 6.5 | 2.2
  DB:Lactate Dehydrogenase AL: number analyzed (Participants) | 93 | 94 | 93 | 92 | 48 | 45
  DB:Lactate Dehydrogenase AL | 0 | 0 | 0 | 0 | 0 | 0
  DB:Lactate Dehydrogenase AH(: number analyzed (Participants) | 93 | 94 | 93 | 92 | 48 | 45
  DB:Lactate Dehydrogenase AH( | 9.7 | 11.7 | 3.2 | 8.7 | 14.6 | 4.4
  F-U:Lactate Dehydrogenase AL: number analyzed (Participants) | 92 | 94 | 90 | 88 | 46 | 45
  F-U:Lactate Dehydrogenase AL | 0 | 0 | 0 | 0 | 0 | 0
  F-U:Lactate Dehydrogenase AH: number analyzed (Participants) | 92 | 94 | 90 | 88 | 46 | 45
  F-U:Lactate Dehydrogenase AH | 6.5 | 7.4 | 7.8 | 9.1 | 13.0 | 6.7
  DB:Serum Protein AL: number analyzed (Participants) | 93 | 96 | 93 | 93 | 48 | 45
  DB:Serum Protein AL | 5.4 | 3.1 | 0 | 0 | 2.1 | 0
  DB:Serum Protein AH: number analyzed (Participants) | 93 | 96 | 93 | 93 | 48 | 45
  DB:Serum Protein AH | 2.2 | 3.1 | 4.3 | 3.2 | 7 | 6.7
  F-U:Serum Protein AL: number analyzed (Participants) | 94 | 94 | 90 | 88 | 46 | 45
  F-U:Serum Protein AL | 0 | 0 | 0 | 0 | 0 | 0
  F-U:Serum Protein AH: number analyzed (Participants) | 94 | 94 | 90 | 88 | 46 | 45
  F-U:Serum Protein AH | 4.3 | 1.1 | 2.2 | 2.3 | 2.2 | 2.2
  DB:Urea Nitrogen AL: number analyzed (Participants) | 93 | 95 | 93 | 93 | 48 | 45
  DB:Urea Nitrogen AL | 6.50 | 0 | 0 | 0 | 0 | 0
  DB:Urea Nitrogen AH: number analyzed (Participants) | 93 | 96 | 93 | 93 | 48 | 45
  DB:Urea Nitrogen AH | 6.5 | 4.2 | 3.2 | 5.4 | 6.3 | 6.7
  F-U:Urea Nitrogen AL: number analyzed (Participants) | 94 | 94 | 90 | 88 | 46 | 45
  F-U:Urea Nitrogen AL | 0 | 0 | 0 | 0 | 0 | 0
  F-U:Urea Nitrogen AH: number analyzed (Participants) | 94 | 94 | 90 | 88 | 46 | 45
  F-U:Urea Nitrogen AH | 6.4 | 4.3 | 2.2 | 1.1 | 8.7 | 0

14. Secondary Outcome: Percentage of Participants With Abnormalities in Clinical Laboratory Tests (Urinalysis)
Description: Percentage of participants with abnormalities in clinical laboratory tests(Urinalysis: abnormally high and low urine granular casts, urine hyaline casts, Urine Leukocytes,Urine Specific Gravity,Urine Squamous Epithelial cell, Urine T.E Cells, Urine Transitinoal erythrocyte count [E.C],Urine Tubular erthrocyte count ) were reported. Abnormality was determined at the investigator's discretion. Participants with abnormally low or high values were reported.
Time Frame: Double blind (DB) phase: Baseline up to Week 48, Follow up (FU) phase: Week 48 up to Week 96
Population: Safety analysis set included all participants who received at least one dose of any of study treatments. Here, 'n' (number analyzed) represents number of participants evaluable at specified categories and "N" (number of participants analyzed) represents number of participants evaluable for this outcome measure. Here 'n=0' signifies no participants were available for analysis at specified timepoint.
Measure: Number; unit: Percentage of participants
Arm/Group | Arm 1: JNJ-73763989 100 mg + JNJ-56136379 250 mg + NA | Arm 2: JNJ-73763989 200 mg + Placebo + NA | Arm 3: JNJ-73763989 100 mg + Placebo + NA | Arm 4: JNJ-73763989 40 mg + Placebo + NA | Arm 5: Placebo + JNJ-56136379 250 mg + NA | Arm 6: Placebo + Placebo + NA
Number analyzed (Participants) | 61 | 61 | 53 | 54 | 29 | 25
Percentage of participants
  DB:Urine Granular Casts AL: number analyzed (Participants) | 1 | 0 | 0 | 1 | 0 | 0
  DB:Urine Granular Casts AL | 0 |  |  | 0 |  |
  DB:Urine Granular Casts AH: number analyzed (Participants) | 1 | 0 | 0 | 1 | 0 | 0
  DB:Urine Granular Casts AH | 100.0 |  |  | 100.0 |  |
  DB:Urine Hyaline Casts AL: number analyzed (Participants) | 3 | 5 | 3 | 4 | 2 | 6
  DB:Urine Hyaline Casts AL | 0 | 0 | 0 | 0 | 0 | 0
  DB:Urine Hyaline Casts AH: number analyzed (Participants) | 3 | 5 | 3 | 4 | 2 | 6
  DB:Urine Hyaline Casts AH | 100.0 | 60.0 | 100.0 | 100.0 | 100.0 | 100.0
  F-U:Urine Hyaline Casts AL: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0
  F-U:Urine Hyaline Casts AL | 0 |  |  |  |  |
  F-U:Urine Hyaline Casts AH: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0
  F-U:Urine Hyaline Casts AH | 100.0 |  |  |  |  |
  DB:Urine Leukocytes AL: number analyzed (Participants) | 47 | 48 | 42 | 39 | 21 | 22
  DB:Urine Leukocytes AL | 0 | 0 | 0 | 0 | 0 | 0
  DB:Urine Leukocytes AH: number analyzed (Participants) | 47 | 48 | 42 | 39 | 21 | 22
  DB:Urine Leukocytes AH | 8.5 | 6.3 | 9.5 | 2.6 | 9.5 | 9.1
  F-U:Urine Leukocytes AL: number analyzed (Participants) | 8 | 7 | 9 | 11 | 4 | 0
  F-U:Urine Leukocytes AL | 0 | 0 | 0 | 0 | 0 |
  F-U:Urine Leukocytes AH: number analyzed (Participants) | 8 | 7 | 9 | 11 | 4 | 0
  F-U:Urine Leukocytes AH | 0 | 0 | 0 | 0 | 25.0 |
  DB:Urine Specific Gravity AL | 1.6 | 0 | 3.8 | 3.7 | 0 | 0
  DB:Urine Specific Gravity AH | 1.6 | 11.5 | 1.9 | 5.6 | 3.4 | 24.0
  F-U:Urine Specific Gravity AL: number analyzed (Participants) | 17 | 15 | 18 | 15 | 8 | 0
  F-U:Urine Specific Gravity AL | 5.9 | 0 | 5.6 | 0 | 0 |
  F-U:Urine Specific Gravity AH: number analyzed (Participants) | 17 | 15 | 18 | 15 | 8 | 0
  F-U:Urine Specific Gravity AH | 5.9 | 0 | 0 | 0 | 0 |
  DB:Urine Squamous Epithelial cell AL: number analyzed (Participants) | 1 | 3 | 4 | 2 | 2 | 2
  DB:Urine Squamous Epithelial cell AL | 0 | 0 | 0 | 0 | 0 | 0
  DB:Urine Squamous Epithelial cellAH: number analyzed (Participants) | 1 | 3 | 4 | 2 | 2 | 2
  DB:Urine Squamous Epithelial cellAH | 100.0 | 66.7 | 75.0 | 50.0 | 50.0 | 50.0
  DB:Urine T.E Cells AL: number analyzed (Participants) | 0 | 1 | 1 | 2 | 1 | 1
  DB:Urine T.E Cells AL |  | 0 | 0 | 0 | 0 | 0
  DB:Urine Transitinoal E.C AH: number analyzed (Participants) | 0 | 1 | 1 | 2 | 1 | 1
  DB:Urine Transitinoal E.C AH |  | 100.0 | 100.0 | 100.0 | 100.0 | 100.0
  DB:Urine Tubular E.C AL: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0
  DB:Urine Tubular E.C AL |  |  |  | 0 |  |
  DB:Urine Tubular E.C AH: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0
  DB:Urine Tubular E.C AH |  |  |  | 100.0 |  |

15. Secondary Outcome: Percentage of Participants With Abnormalities in Electrocardiogram (ECG)
Description: Percentage of participants with abnormalities in ECG parameters (heart rate, PR interval, QRS duration, and QTcF interval) were reported. Abnormality criteria: Heart rate abnormally low (AL): <45 beats per minute (bpm); PR interval AH:>220 msec; QRS duration AH:>120 msec; QTcF borderline prolonged (BP) QT: 450 msec to <=480 msec. Participants with abnormally low or high values were reported.
Time Frame: Double blind (DB) phase: Baseline (Day 1) up to Week 48, Follow up (FU) phase: Week 48 up to Week 96
Population: Safety analysis set included all participants who received at least one dose of any of the study treatments. Here, 'N' (number of participant analysed) signifies number of participant who were evaluable for this outcome measure and 'n' (number analyzed) represents number of participant evaluable for specified categories.
Measure: Number; unit: Percentage of participants
Arm/Group | Arm 1: JNJ-73763989 100 mg + JNJ-56136379 250 mg + NA | Arm 2: JNJ-73763989 200 mg + Placebo + NA | Arm 3: JNJ-73763989 100 mg + Placebo + NA | Arm 4: JNJ-73763989 40 mg + Placebo + NA | Arm 5: Placebo + JNJ-56136379 250 mg + NA | Arm 6: Placebo + Placebo + NA
Number analyzed (Participants) | 93 | 95 | 91 | 92 | 47 | 45
Percentage of participants
  DB Phase: Heart Rate AL | 0 | 2.1 | 1.1 | 3.3 | 0 | 0
  FU Phase: Heart Rate AL: number analyzed (Participants) | 92 | 84 | 83 | 84 | 46 | 1
  FU Phase: Heart Rate AL | 0 | 0 | 0 | 0 | 2.2 | 0
  DB Phase: PR interval AH | 1.1 | 0 | 3.3 | 1.1 | 4.3 | 2.2
  FU Phase: PR interval AH: number analyzed (Participants) | 92 | 84 | 83 | 84 | 46 | 1
  FU Phase: PR interval AH | 0 | 0 | 1.2 | 0 | 0 | 0
  DB Phase: QRS duration AH | 2.2 | 1.1 | 1.1 | 0 | 0 | 2.2
  FU Phase: QRS duration AH: number analyzed (Participants) | 92 | 84 | 83 | 84 | 46 | 1
  FU Phase: QRS duration AH | 2.2 | 0 | 0 | 0 | 0 | 0
  DB Phase: QTcF interval BP-QT | 2.2 | 2.1 | 3.3 | 1.1 | 0 | 2.2
  FU Phase: QTcF interval BP-QT: number analyzed (Participants) | 92 | 84 | 83 | 84 | 46 | 1
  FU Phase: QTcF interval BP-QT | 1.1 | 0 | 2.4 | 1.2 | 0 | 0

16. Secondary Outcome: Percentage of Participants With Abnormalities in Vital Signs
Description: Percentage of participants with abnormalities in vital signs parameters (pulse rate, diastolic and systolic blood pressure) were reported. Abnormality criteria: Pulse rate AL:<=45 bpm; Systolic blood pressure (SBP) AL: <=90 millimeters of mercury (mmHg), mild:>140 mmHg to <160 mmHg; moderate:>=160 mmHg to <180 mmHg; Diastolic blood pressure (DBP): AL: <=150 mmHg; mild:>90 mmHg to <100 mmHg; moderate: >=100 mmHg to <110 mmHg; severe:>=110 mmHg. Abnormality was determined at the investigator's discretion. Participants with abnormally low or high values were reported.
Time Frame: Double blind (DB) phase: Baseline (Day 1) up to Week 48, Follow up (FU) phase: Week 48 up to Week 96
Population: Safety analysis set included all participants who received at least one dose of any of the study treatments. Here, 'N' (number of subject analysed) signifies number of participants who were evaluable for this outcome measure and 'n' (number analyzed) represented number of participants evaluable for the specified categories.
Measure: Number; unit: Percentage of participants
Arm/Group | Arm 1: JNJ-73763989 100 mg + JNJ-56136379 250 mg + NA | Arm 2: JNJ-73763989 200 mg + Placebo + NA | Arm 3: JNJ-73763989 100 mg + Placebo + NA | Arm 4: JNJ-73763989 40 mg + Placebo + NA | Arm 5: Placebo + JNJ-56136379 250 mg + NA | Arm 6: Placebo + Placebo + NA
Number analyzed (Participants) | 94 | 96 | 93 | 93 | 48 | 45
Percentage of participants
  DB:Pulse rate AL: number analyzed (Participants) | 93 | 96 | 93 | 93 | 48 | 45
  DB:Pulse rate AL | 1.1 | 4.2 | 2.2 | 2.2 | 0 | 0
  DB:Pulse rate AH: number analyzed (Participants) | 93 | 96 | 93 | 93 | 48 | 45
  DB:Pulse rate AH | 0 | 2.1 | 1.1 | 2.2 | 0 | 0
  FU:Pulse rate AL: number analyzed (Participants) | 94 | 94 | 90 | 88 | 46 | 45
  FU:Pulse rate AL | 1.1 | 0 | 1.1 | 2.3 | 0 | 0
  FU:Pulse rate AH: number analyzed (Participants) | 94 | 94 | 90 | 88 | 46 | 45
  FU:Pulse rate AH | 0 | 0 | 0 | 1.1 | 0 | 0
  DB: DBP AL: number analyzed (Participants) | 93 | 96 | 93 | 93 | 48 | 45
  DB: DBP AL | 4.3 | 1.0 | 4.3 | 4.3 | 0 | 2.2
  DB: DBP mild: number analyzed (Participants) | 93 | 96 | 93 | 93 | 48 | 45
  DB: DBP mild | 20.4 | 18.8 | 12.9 | 14.0 | 0 | 6.7
  DB: DBP moderate: number analyzed (Participants) | 93 | 96 | 93 | 93 | 48 | 45
  DB: DBP moderate | 4.3 | 4.2 | 3.2 | 3.2 | 0 | 0
  DB: DBP severe: number analyzed (Participants) | 93 | 96 | 93 | 93 | 48 | 45
  DB: DBP severe | 0 | 0 | 0 | 1.1 | 0 | 0
  FU: DBP AL: number analyzed (Participants) | 94 | 94 | 90 | 88 | 46 | 45
  FU: DBP AL | 1.1 | 1.1 | 0 | 1.1 | 0 | 0
  FU: DBP mild: number analyzed (Participants) | 94 | 94 | 90 | 88 | 46 | 45
  FU: DBP mild | 10.16 | 10.16 | 4.4 | 12.5 | 0 | 8.9
  FU: DBP moderate: number analyzed (Participants) | 94 | 94 | 90 | 88 | 46 | 45
  FU: DBP moderate | 1.1 | 2.1 | 4.4 | 1.1 | 0 | 0
  DB: SBP AL: number analyzed (Participants) | 93 | 96 | 93 | 93 | 48 | 45
  DB: SBP AL | 0 | 6.3 | 2.2 | 6.5 | 0 | 4.4
  DB: SBP mild: number analyzed (Participants) | 93 | 96 | 93 | 93 | 48 | 45
  DB: SBP mild | 23.7 | 18.8 | 12.9 | 22.6 | 0 | 17.8
  DB: SBP moderate: number analyzed (Participants) | 93 | 96 | 93 | 93 | 48 | 45
  DB: SBP moderate | 4.3 | 3.1 | 4.3 | 2.2 | 0 | 2.2
  FU: SBP AL: number analyzed (Participants) | 94 | 94 | 90 | 88 | 46 | 45
  FU: SBP AL | 3.2 | 2.1 | 1.1 | 4.5 | 0 | 0
  FU: SBP mild: number analyzed (Participants) | 94 | 94 | 90 | 88 | 46 | 45
  FU: SBP mild | 12.8 | 12.8 | 11.1 | 10.2 | 0 | 4.4
  FU: SBP moderate: number analyzed (Participants) | 94 | 94 | 90 | 88 | 46 | 45
  FU: SBP moderate | 0 | 2.1 | 2.2 | 2.1 | 0 | 0

17. Secondary Outcome: Percentage of Participants With HBsAg Seroclearance 24 Weeks After Completion of All Study Intervention at Week 48
Description: Percentage of participants with HBsAg seroclearance 24 weeks after completion of all study intervention at Week 48 were reported. HBsAg seroclearance was defined as HBsAg (less than [<] lower limit of quantification LLOQ [0.05 IU/mL]). Responder was defined as a participant who achieved functional cure at Week 72. A participant was defined as having achieved functional cure at Week 72 if he/she: had met the criteria for stopping NA treatment at Week 48 and stopped treatment; had HBsAg seroclearance at Week 72 (that is, 24 weeks after stopping all study interventions); did not require NA re-treatment between Weeks 48 and 72. Multiple Imputation using a longitudinal multiple regression model was applied to impute missing data.
Time Frame: Week 72
Population: mITT set was defined as all participants who were randomized in the study and received at least one dose of study treatment excluding those participants impacted by the COVID-19 pandemic defined as those participants who, because of COVID-19 or similar pandemic-related reasons, withdrew prematurely from the study prior to Week 44, or had no efficacy assessment for the primary outcome measure.
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm 1: JNJ-73763989 100 mg + JNJ-56136379 250 mg + NA | Arm 2: JNJ-73763989 200 mg + Placebo + NA | Arm 3: JNJ-73763989 100 mg + Placebo + NA | Arm 4: JNJ-73763989 40 mg + Placebo + NA | Arm 5: Placebo + JNJ-56136379 250 mg + NA | Arm 6: Placebo + Placebo + NA
Number analyzed (Participants) | 94 | 94 | 92 | 91 | 48 | 45
Percentage of participants | 0.0 [0.00 to 3.14] | 0.0 [0.00 to 3.14] | 0.0 [0.00 to 3.20] | 0.0 [0.00 to 3.24] | 0.0 [0.00 to 6.05] | 2.2 [0.11 to 10.11]

18. Secondary Outcome: Percentage of Participants With HBsAg Seroclearance 48 Weeks After Completion of All Study Intervention at Week 48
Description: Percentage of participants with HBsAg seroclearance 48 weeks after completion of all study intervention at Week 48 were reported. HBsAg Seroclearance was defined as HBsAg <LLOQ (0.05 IU/mL). A responder was defined as a participant who achieved HBsAg seroclearance at Week 96 if the participant completed 48 weeks of treatment, met the criteria for stopping NA treatment at Week 48, did not require NA re-treatment between Week 48 and Week 96, and had HBsAg seroclearance at Week 96. Multiple Imputation using a longitudinal multiple regression model was applied to impute missing data.
Time Frame: Week 96
Population: mITT analysis set included all participants who were randomized in the study and received at least one dose of study treatment excluding those participants impacted by the pandemic defined as those participants who, because of COVID-19 or similar pandemics related reasons, withdrew prematurely from the study prior to Week 44.
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm 1: JNJ-73763989 100 mg + JNJ-56136379 250 mg + NA | Arm 2: JNJ-73763989 200 mg + Placebo + NA | Arm 3: JNJ-73763989 100 mg + Placebo + NA | Arm 4: JNJ-73763989 40 mg + Placebo + NA | Arm 5: Placebo + JNJ-56136379 250 mg + NA | Arm 6: Placebo + Placebo + NA
Number analyzed (Participants) | 94 | 94 | 92 | 91 | 48 | 45
Percentage of participants | 0.0 (0.00) [0.00 to 3.14] | 1.1 (0.05) [0.05 to 4.95] | 0.0 (0.00) [0.00 to 3.20] | 0.0 (0.00) [0.00 to 3.24] | 0.0 (0.00) [0.00 to 6.05] | 2.2 (0.11) [0.11 to 10.11]

19. Secondary Outcome: Percentage of Participants With HBV DNA <LLOQ 24 and 48 Weeks After Completion of All Study Intervention at Week 48
Description: Percentage of participants with HBV DNA <LLOQ at 24 and 48 weeks after completion of all study intervention at Week 48 were reported. A responder was defined as a participant who achieved HBV DNA <LLOQ 24 and 48 weeks after stopping all study treatments at any time during the study and without restarting NA treatment thereafter.
Time Frame: Weeks 72 and 96
Population: mITT analysis set: all participants who were randomized in study and received at least one dose of study treatment excluding those participants impacted by pandemic: those participants who, because of COVID-19 or similar pandemics related reasons, withdrew prematurely from study prior to Week 44. Here, 'n' (number analyzed) represents participants evaluable at the specified timepoint.
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm 1: JNJ-73763989 100 mg + JNJ-56136379 250 mg + NA | Arm 2: JNJ-73763989 200 mg + Placebo + NA | Arm 3: JNJ-73763989 100 mg + Placebo + NA | Arm 4: JNJ-73763989 40 mg + Placebo + NA | Arm 5: Placebo + JNJ-56136379 250 mg + NA | Arm 6: Placebo + Placebo + NA
Number analyzed (Participants) | 94 | 94 | 92 | 91 | 48 | 45
Percentage of participants
  Week 72 | 5.3 [2.12 to 10.86] | 16.0 [10.10 to 23.50] | 7.6 [3.63 to 13.82] | 1.1 [0.06 to 5.11] | 0.0 [0.00 to 6.05] | 4.4 [0.80 to 13.34]
  Week 96 | 6.4 [2.82 to 12.21] | 9.6 [5.09 to 16.11] | 5.4 [2.17 to 11.09] | 1.1 [0.06 to 5.11] | 2.1 [0.11 to 9.51] | 0.0 [0.00 to 6.44]

20. Secondary Outcome: Percentage of Participants Meeting the NA Treatment Completion Criteria During Follow-up
Description: Percentage of participants meeting the NA treatment completion criteria during follow-up were reported. A participant was defined as a responder in meeting the NA treatment completion criteria at Week 48, if the following criteria were met based on the clinical laboratory tests performed at Week 44: participants had alanine transaminase (ALT) less than (<) 3*upper limit of normal range (ULN); had hepatitis B virus deoxyribonucleic acid (HBV DNA) < lower limit of quantification (LLOQ); was hepatitis B e antigen (HBeAg)-negative; had hepatitis B surface antigen (HBsAg) <10 international units per milliliter (IU/mL). A responder was defined as a participant who stopped NA at Week 48 and met the NA treatment completion criteria at any time during the follow-up phase, regardless of the treatment duration.
Time Frame: Week 48 up to Week 96
Population: mITT analysis set included all participants who were randomised in the study and received at least one dose of study treatment excluding those participants impacted by the pandemic defined as those subjects who, because of COVID-19 or similar pandemics related reasons, withdrew prematurely from the study prior to Week 44.
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm 1: JNJ-73763989 100 mg + JNJ-56136379 250 mg + NA | Arm 2: JNJ-73763989 200 mg + Placebo + NA | Arm 3: JNJ-73763989 100 mg + Placebo + NA | Arm 4: JNJ-73763989 40 mg + Placebo + NA | Arm 5: Placebo + JNJ-56136379 250 mg + NA | Arm 6: Placebo + Placebo + NA
Number analyzed (Participants) | 94 | 94 | 92 | 91 | 48 | 45
Percentage of participants | 11.7 [6.70 to 18.63] | 27.7 [20.16 to 36.25] | 16.3 [10.33 to 23.99] | 4.4 [1.52 to 9.78] | 0.0 [0.00 to 6.05] | 2.2 [0.11 to 10.11]

21. Secondary Outcome: Percentage of Participants With HBsAg Seroclearance After Completion of NA Treatment at Weeks 60, 84, and 96
Description: Percentage of participants with HBsAg seroclearance after completion of NA treatment at Weeks 60, 84, and 96 were reported. Seroclearance of HBsAg was defined as HBsAg level <LLOQ (0.05 IU/mL). For Week 60: a responder was defined as a participant who achieved HBsAg seroclearance 12 weeks off treatment if the subject achieved HBsAg seroclearance 12 weeks after stopping; for Week 84:A responder was defined as a participant who achieved HBsAg seroclearance 36 weeks off-treatment if the participant achieved HBsAg seroclearance 36 weeks after stopping all study treatments; for Week 96:A responder was defined as a participant who achieved HBsAg seroclearance at Week 96 if the participant completed 48 weeks of treatment, met the criteria for stopping NA treatment at Week 48, did not require NA re-treatment between Week 48 and Week 96, and had HBsAg seroclearance at Week 96.
Time Frame: Weeks 60, 84, and 96
Population: as for outcome 19
Measure: Number (90% Confidence Interval); unit: Percentage of of participants
Arm/Group | Arm 1: JNJ-73763989 100 mg + JNJ-56136379 250 mg + NA | Arm 2: JNJ-73763989 200 mg + Placebo + NA | Arm 3: JNJ-73763989 100 mg + Placebo + NA | Arm 4: JNJ-73763989 40 mg + Placebo + NA | Arm 5: Placebo + JNJ-56136379 250 mg + NA | Arm 6: Placebo + Placebo + NA
Number analyzed (Participants) | 94 | 94 | 92 | 91 | 48 | 45
Percentage of of participants
  Week 60: number analyzed (Participants) | 9 | 22 | 18 | 5 | 0 | 1
  Week 60 | 0.0 [0.00 to 28.31] | 9.1 [1.64 to 25.95] | 0.0 [0.00 to 15.33] | 0.0 [0.00 to 45.07] |  | 0.0 [0.00 to 95.00]
  Week 84: number analyzed (Participants) | 10 | 22 | 14 | 5 | 0 | 1
  Week 84 | 0.0 [0.00 to 25.89] | 9.1 [1.64 to 25.95] | 0.0 [0.00 to 19.26] | 0.0 [0.00 to 45.07] |  | 100.0 [5.0 to 100.0]
  Week 96 | 0.0 [0.00 to 3.14] | 1.1 [0.05 to 4.95] | 0.0 [0.00 to 3.20] | 0.0 [0.00 to 3.24] | 0.0 [0.00 to 6.05] | 2.2 [0.11 to 10.11]

22. Secondary Outcome: Percentage of Participants Who Required NA Re-treatment During Follow-up
Description: Percentage of participants who required NA re-treatment during follow-up were reported. Responder was defined as a participant who met the criteria for NA re-treatment at any time during follow-up, for those participants who met the NA treatment completion criteria at any time during the study and actually stopped NA treatment. NA re-treatment criteria: (1) Re-start NA treatment immediately with signs of decreasing liver function based on laboratory findings (eg, International Normalized Ratio [INR], direct bilirubin) or clinical assessment (eg, ascites, hepatic encephalopathy). (2) Immediately with an HBV DNA value of >100,000 IU/mL (irrespective of confirmation and/or ALT increase). (3) With confirmed post-treatment HBeAg seroreversion (HBeAg positive after it was negative at NA completion) (4) With confirmed* post-treatment increases in HBV DNA >2,000 IU/mL and ALT >5x ULN (5) With confirmed* post-treatment increases in HBV DNA >20,000 IU/mL.
Time Frame: Week 48 up to Week 96
Population: mITT analysis set included all participants who were randomised in the study and received at least one dose of study treatment excluding those participant impacted by the pandemic defined as those participant who, because of COVID-19 or similar pandemics related reasons, withdrew prematurely from the study prior to Week 44.
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm 1: JNJ-73763989 100 mg + JNJ-56136379 250 mg + NA | Arm 2: JNJ-73763989 200 mg + Placebo + NA | Arm 3: JNJ-73763989 100 mg + Placebo + NA | Arm 4: JNJ-73763989 40 mg + Placebo + NA | Arm 5: Placebo + JNJ-56136379 250 mg + NA | Arm 6: Placebo + Placebo + NA
Number analyzed (Participants) | 94 | 94 | 92 | 91 | 48 | 45
Percentage of participants | 1.1 (0.05) [0.05 to 4.95] | 1.1 (0.05) [0.05 to 4.95] | 2.2 (0.39) [0.39 to 6.69] | 0.0 (0.00) [0.00 to 3.24] | 0.0 (0.00) [0.00 to 6.05] | 0.0 (0.00) [0.00 to 6.44]

23. Secondary Outcome: Percentage of Participants With Flares
Description: Percentage of participants with flares (virologic, biochemical, and clinical) were reported. Virologic flare: confirmed HBV DNA >peak threshold ( 20,000 IU/mL 2,000 IU/mL and 200 IU/mL); biochemical Flare: confirmed ALT and/or AST increase of 3*ULN and 3*nadir; clinical flare: confirmed HBV DNA >peak threshold and confirmed ALT and/or AST increase of 3*ULN and 3*nadir. Virologic and clinical flare was assessed only for those participants who were off-treatment and had HBV DNA<LLOQ at the last observed time point on all study treatments and biochemical flares was identified on treatment and off treatment, respectively. Each virologic flare was categorized based on the confirmed (i.e., two consecutive values) peak HBV DNA above any of the three thresholds within the start and end date of that flare as follows: 20,000 IU/mL 2,000 IU/mL and 200 IU/mL. A participant was defined as off-treatment failure if he/she required NA re-treatment after stopping all study interventions.
Time Frame: Follow-up phase (Week 48 up to Week 96)
Population: mITT analysis set included all participants who were randomised in the study and received at least one dose of study treatment excluding those participants impacted by the pandemic defined as those participants who, because of COVID-19 or similar pandemics related reasons, withdrew prematurely from the study prior to Week 44. Here, 'n' (number analysed) represents number of participants evaluable for the specified categories.
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm 1: JNJ-73763989 100 mg + JNJ-56136379 250 mg + NA | Arm 2: JNJ-73763989 200 mg + Placebo + NA | Arm 3: JNJ-73763989 100 mg + Placebo + NA | Arm 4: JNJ-73763989 40 mg + Placebo + NA | Arm 5: Placebo + JNJ-56136379 250 mg + NA | Arm 6: Placebo + Placebo + NA
Number analyzed (Participants) | 94 | 94 | 92 | 91 | 48 | 45
Percentage of participants
  Biochemical: On NA | 0.0 [0.00 to 3.14] | 0.0 [0.00 to 3.14] | 0.0 [0.00 to 3.20] | 0.0 [0.00 to 3.24] | 2.1 [0.11 to 9.51] | 0.0 [0.00 to 6.44]
  Biochemical: Off NA: number analyzed (Participants) | 33 | 40 | 40 | 18 | 10 | 10
  Biochemical: Off NA | 0.0 [0.00 to 8.68] | 2.5 [1.13 to 11.32] | 0.0 [0.00 to 7.22] | 0.0 [0.00 to 14.59] | 0.0 [0.00 to 25.89] | 0.0 [0.00 to 25.89]
  Virologic HBVDNA>200:Off NA: number analyzed (Participants) | 30 | 37 | 37 | 14 | 9 | 10
  Virologic HBVDNA>200:Off NA | 13.3 [4.69 to 27.96] | 24.3 [13.32 to 38.61] | 21.6 [11.24 to 35.64] | 14.3 [2.60 to 38.54] | 0.0 [0.00 to 28.31] | 0.0 [0.00 to 25.89]
  Virologic HBVDNA>2000:Off NA: number analyzed (Participants) | 30 | 37 | 37 | 14 | 9 | 10
  Virologic HBVDNA>2000:Off NA | 3.3 [0.17 to 14.86] | 2.7 [0.14 to 12.19] | 8.1 [2.25 to 19.64] | 7.1 [0.37 to 29.67] | 0.0 [0.00 to 28.21] | 10.0 [0.51 to 39.42]
  Virologic HBVDNA>20000:Off NA: number analyzed (Participants) | 30 | 37 | 37 | 14 | 9 | 10
  Virologic HBVDNA>20000:Off NA | 3.0 [0.17 to 14.86] | 2.7 [0.14 to 12.19] | 5.4 [0.97 to 16.05] | 0.0 [0.00 to 19.26] | 0.0 [0.00 to 8.31] | 0.0 [0.00 to 25.89]
  Clinical HBVDNA>200:Off NA: number analyzed (Participants) | 30 | 37 | 37 | 14 | 9 | 10
  Clinical HBVDNA>200:Off NA | 0.0 [0.00 to 9.50] | 0.0 [0.00 to 7.78] | 0.0 [0.00 to 7.78] | 0.0 [0.00 to 19.26] | 0.0 [0.00 to 28.31] | 0.0 [0.00 to 25.89]
  Clinical HBVDNA>2000:Off NA: number analyzed (Participants) | 30 | 37 | 37 | 14 | 9 | 10
  Clinical HBVDNA>2000:Off NA | 0.0 [0.00 to 9.50] | 0.0 [0.00 to 7.78] | 0.0 [0.00 to 7.78] | 0.0 [0.00 to 19.26] | 0.0 [0.00 to 28.31] | 0.0 [0.00 to 25.89]
  Clinical HBVDNA>20000:Off NA: number analyzed (Participants) | 30 | 37 | 14 | 9 | 10 | 10
  Clinical HBVDNA>20000:Off NA | 0.0 [0.00 to 9.50] | 2.7 [0.14 to 12.19] | 0.0 [0.00 to 7.78] | 0.0 [0.00 to 19.26] | 0.0 [0.00 to 28.31] | 0.0 [0.00 to 25.89]

24. Secondary Outcome: Number of Participants With (Sustained) Reduction, Suppression, and/or Seroclearance Considering Single and Multiple Marker
Description: Number of participants with (sustained) reduction considering multiple markers were reported. HBV DNA results <LLOQ were reported as: (a) target detected, that is, traces of HBV DNA were detected/found but were too low to be quantified, or (b) target not detected, that is, no traces of HBV DNA were detected/found. LLOQ value for HBV DNA was 20 IU/mL.
Time Frame: Weeks 12, 24, 36 and 48
Population: mITT population. Here, 'N' (number of participants analyzed) signifies number of participants with non-missing data for both blood markers at specified time point after stopping all study treatments (including NA), who also met NA treatment completion criteria and at least 24 week off-treatment data available; and 'n' (number analysed) represents number of participants evaluable at specified timepoints.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: JNJ-73763989 100 mg + JNJ-56136379 250 mg + NA | Arm 2: JNJ-73763989 200 mg + Placebo + NA | Arm 3: JNJ-73763989 100 mg + Placebo + NA | Arm 4: JNJ-73763989 40 mg + Placebo + NA | Arm 5: Placebo + JNJ-56136379 250 mg + NA | Arm 6: Placebo + Placebo + NA
Number analyzed (Participants) | 10 | 25 | 18 | 5 | 1 | 1
Participants
  Week 12: HBsAg < LLOQ and HBV DNA < LLOQ for target detected and not detected: number analyzed (Participants) | 10 | 25 | 17 | 5 | 1 | 1
  Week 12: HBsAg < LLOQ and HBV DNA < LLOQ for target detected and not detected | 0 | 1 | 0 | 0 | 0 | 0
  Week 12: HBsAg >= LLOQ and HBV DNA < LLOQ for target detected and not detected: number analyzed (Participants) | 10 | 25 | 17 | 5 | 1 | 1
  Week 12: HBsAg >= LLOQ and HBV DNA < LLOQ for target detected and not detected | 6 | 20 | 7 | 2 | 1 | 0
  Week 24: HBsAg < LLOQ and HBV DNA < LLOQ for target detected and not detected: number analyzed (Participants) | 10 | 24 | 16 | 5 | 1 | 1
  Week 24: HBsAg < LLOQ and HBV DNA < LLOQ for target detected and not detected | 0 | 1 | 0 | 0 | 0 | 1
  Week 24: HBsAg >= LLOQ and HBV DNA < LLOQ for target detected and not detected: number analyzed (Participants) | 10 | 24 | 16 | 5 | 1 | 1
  Week 24: HBsAg >= LLOQ and HBV DNA < LLOQ for target detected and not detected | 4 | 13 | 6 | 1 | 1 | 0
  Week 36: HBsAg < LLOQ and HBV DNA < LLOQ for target detected and not detected: number analyzed (Participants) | 9 | 23 | 18 | 5 | 1 | 1
  Week 36: HBsAg < LLOQ and HBV DNA < LLOQ for target detected and not detected | 0 | 2 | 0 | 0 | 0 | 1
  Week 36: HBsAg >= LLOQ and HBV DNA < LLOQ for target detected and not detected: number analyzed (Participants) | 9 | 23 | 18 | 5 | 1 | 1
  Week 36: HBsAg >= LLOQ and HBV DNA < LLOQ for target detected and not detected | 3 | 8 | 7 | 2 | 1 | 0
  Week 48: HBsAg < LLOQ and HBV DNA < LLOQ for target detected and not detected: number analyzed (Participants) | 10 | 23 | 18 | 5 | 1 | 1
  Week 48: HBsAg < LLOQ and HBV DNA < LLOQ for target detected and not detected | 0 | 1 | 0 | 0 | 0 | 0
  Week 48: HBsAg >= LLOQ and HBV DNA < LLOQ for target detected and not detected: number analyzed (Participants) | 10 | 23 | 18 | 5 | 1 | 1
  Week 48: HBsAg >= LLOQ and HBV DNA < LLOQ for target detected and not detected | 6 | 7 | 5 | 1 | 1 | 0

25. Secondary Outcome: Percentage of Participants With HBsAg Seroconversion
Description: HBsAg seroconversion was defined as achieving HBsAg seroclearance (HBsAg [quantitative] <LLOQ [0.05 IU/mL]) together with an appearance of anti-HBs antibodies (baseline anti-HBs antibodies [quantitative] <LLOQ and a post-baseline assessment greater than or equal to [>=] LLOQ).
Time Frame: Weeks 48, 60, 72, and 96
Population: mITT analysis set: all participants who were randomized in study and received at least one dose of study treatment excluding those participants impacted by pandemic: those participants who, because of COVID-19 or similar pandemics related reasons, withdrew prematurely from study prior to Week 44. Here, 'N' (number of participants analyzed) signifies participants who were evaluable for this outcome measure and 'n' (number analyzed) represents participants evaluable at the specified timepoint.
Measure: Number; unit: Percentage of participants
Arm/Group | Arm 1: JNJ-73763989 100 mg + JNJ-56136379 250 mg + NA | Arm 2: JNJ-73763989 200 mg + Placebo + NA | Arm 3: JNJ-73763989 100 mg + Placebo + NA | Arm 4: JNJ-73763989 40 mg + Placebo + NA | Arm 5: Placebo + JNJ-56136379 250 mg + NA | Arm 6: Placebo + Placebo + NA
Number analyzed (Participants) | 87 | 89 | 83 | 85 | 45 | 42
Percentage of participants
  Week 48: number analyzed (Participants) | 86 | 89 | 83 | 85 | 44 | 42
  Week 48 | 0.0 | 1.1 | 0.0 | 0.0 | 0.0 | 0.0
  Week 60: number analyzed (Participants) | 85 | 83 | 78 | 81 | 45 | 41
  Week 60 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Week 72: number analyzed (Participants) | 83 | 82 | 76 | 82 | 45 | 42
  Week 72 | 0.0 | 0.0 | 1.3 | 0.0 | 0.0 | 2.4
  Week 96: number analyzed (Participants) | 87 | 81 | 80 | 80 | 42 | 42
  Week 96 | 0.0 | 1.2 | 0.0 | 0.0 | 0.0 | 0.0

26. Secondary Outcome: Percentage of Participants With HBeAg Seroconversion
Description: HBeAg seroconversion was defined as achieving HBeAg seroclearance (HBeAg [quantitative] <LLOQ) together with an appearance of anti-HBe antibodies (baseline anti-HBe antibodies [qualitative] with a "negative" result and a post-baseline assessment with "positive" result.
Time Frame: Weeks 48, 60, 72, and 96
Population: mITT population. Here, 'N' (number of participants analyzed) signifies HbeAg positive participants who were evaluable for this outcome measure and 'n' (number analyzed) represents participants evaluable at the specified timepoint.
Measure: Number; unit: Percentage of participants
Arm/Group | Arm 1: JNJ-73763989 100 mg + JNJ-56136379 250 mg + NA | Arm 2: JNJ-73763989 200 mg + Placebo + NA | Arm 3: JNJ-73763989 100 mg + Placebo + NA | Arm 4: JNJ-73763989 40 mg + Placebo + NA | Arm 5: Placebo + JNJ-56136379 250 mg + NA | Arm 6: Placebo + Placebo + NA
Number analyzed (Participants) | 25 | 28 | 23 | 25 | 14 | 11
Percentage of participants
  Week 48: number analyzed (Participants) | 25 | 28 | 23 | 24 | 13 | 11
  Week 48 | 4.0 | 3.6 | 8.7 | 0 | 0 | 18.2
  Week 60: number analyzed (Participants) | 25 | 27 | 22 | 23 | 14 | 10
  Week 60 | 4.3 | 7.4 | 4.5 | 0 | 0 | 20.0
  Week 72: number analyzed (Participants) | 24 | 27 | 22 | 25 | 14 | 11
  Week 72 | 4.2 | 3.7 | 9.1 | 0 | 0 | 18.2
  Week 96: number analyzed (Participants) | 25 | 27 | 23 | 24 | 13 | 11
  Week 96 | 8.0 | 14.8 | 13.0 | 4.2 | 7.7 | 18.2

27. Secondary Outcome: Change From Baseline in HBsAg Levels
Description: Change from baseline in HBsAg levels was reported.
Time Frame: Baseline, Weeks 12, 24, 48, 60, 72, 96
Population: mITT analysis set included all participants who were randomized in the study and received at least one dose of study treatment excluding those participants impacted by the pandemic defined as those participants who, because of COVID-19 or similar pandemics related reasons, withdrew prematurely from the study prior to Week 44. Here, 'n' (number analyzed) represents number of participants evaluable for the specified timepoints.
Measure: Mean (Standard Deviation); unit: Log10 international units per milliliter
Arm/Group | Arm 1: JNJ-73763989 100 mg + JNJ-56136379 250 mg + NA | Arm 2: JNJ-73763989 200 mg + Placebo + NA | Arm 3: JNJ-73763989 100 mg + Placebo + NA | Arm 4: JNJ-73763989 40 mg + Placebo + NA | Arm 5: Placebo + JNJ-56136379 250 mg + NA | Arm 6: Placebo + Placebo + NA
Number analyzed (Participants) | 94 | 94 | 92 | 91 | 48 | 45
Log10 international units per milliliter
  Baseline | 3.66 (0.691) | 3.83 (0.721) | 3.70 (0.778) | 3.81 (0.678) | 3.63 (0.681) | 3.83 (0.714)
  Week 12: number analyzed (Participants) | 92 | 92 | 86 | 88 | 45 | 45
  Week 12 | -0.96 (0.533) | -1.51 (0.790) | -1.24 (0.646) | -0.82 (0.361) | -0.01 (0.286) | -0.07 (0.244)
  Week 24: number analyzed (Participants) | 91 | 92 | 88 | 88 | 45 | 44
  Week 24 | -1.52 (0.582) | -2.22 (0.768) | -1.84 (0.612) | -1.26 (0.430) | -0.05 (0.356) | -0.12 (0.350)
  Week 48: number analyzed (Participants) | 87 | 91 | 88 | 86 | 45 | 44
  Week 48 | -1.76 (0.643) | -2.58 (0.996) | -2.09 (0.665) | -1.50 (0.470) | -0.07 (0.354) | -0.22 (0.854)
  Week 60: number analyzed (Participants) | 87 | 85 | 84 | 83 | 46 | 1
  Week 60 | -1.59 (0.613) | -2.21 (0.975) | -1.75 (0.699) | -1.22 (0.456) | -0.12 (0.367) | -0.21 (0.747)
  Week 72: number analyzed (Participants) | 85 | 83 | 82 | 84 | 46 | 45
  Week 72 | -1.38 (0.630) | -1.85 (0.927) | -1.50 (0.783) | -1.01 (0.487) | -0.15 (0.366) | -0.26 (1.032)
  Week 96: number analyzed (Participants) | 89 | 82 | 85 | 82 | 44 | 45
  Week 96 | -1.04 (0.634) | -1.39 (0.895) | -1.15 (0.744) | -0.74 (0.497) | -0.14 (0.360) | -0.25 (1.031)

28. Secondary Outcome: Change From Baseline in HBeAg Levels
Description: Change from baseline in HBeAg levels was reported.
Time Frame: Baseline, Weeks 12, 24, 48, 60, 72, 96
Population: mITT analysis set: all HbeAg + participants who were randomized in study and received at least one dose of study treatment excluding those participants impacted by pandemic: those participants who, because of COVID-19 or similar pandemics related reasons, withdrew prematurely from study prior to Week 44. Here, 'n' (number analyzed) represents participants evaluable at the specified timepoint.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | Arm 1: JNJ-73763989 100 mg + JNJ-56136379 250 mg + NA | Arm 2: JNJ-73763989 200 mg + Placebo + NA | Arm 3: JNJ-73763989 100 mg + Placebo + NA | Arm 4: JNJ-73763989 40 mg + Placebo + NA | Arm 5: Placebo + JNJ-56136379 250 mg + NA | Arm 6: Placebo + Placebo + NA
Number analyzed (Participants) | 27 | 30 | 25 | 30 | 15 | 13
log10 IU/mL
  Baseline | 1.22 (1.494) | 1.60 (1.449) | 1.68 (1.540) | 1.26 (1.318) | 0.81 (1.261) | 1.03 (1.435)
  Week 12: number analyzed (Participants) | 27 | 27 | 23 | 29 | 13 | 10
  Week 12 | -0.82 (0.746) | -0.90 (0.629) | -0.95 (0.502) | -0.44 (0.273) | -0.60 (0.652) | -0.32 (0.425)
  Week 24: number analyzed (Participants) | 27 | 29 | 25 | 30 | 13 | 13
  Week 24 | -1.00 (0.880) | -1.17 (0.832) | -1.12 (0.636) | -0.54 (0.372) | -0.77 (0.817) | -0.59 (0.782)
  Week 48: number analyzed (Participants) | 26 | 28 | 24 | 27 | 14 | 13
  Week 48 | -1.43 (1.194) | -1.50 (1.142) | -1.53 (0.999) | -0.78 (0.550) | -0.84 (0.876) | -0.96 (1.325)
  Week 60: number analyzed (Participants) | 25 | 27 | 24 | 27 | 15 | 12
  Week 60 | -1.40 (1.253) | -1.61 (1.168) | -1.32 (0.763) | -0.83 (0.600) | -0.87 (0.874) | -1.03 (1.384)
  Week 72: number analyzed (Participants) | 25 | 27 | 23 | 28 | 15 | 13
  Week 72 | -1.50 (1.276) | -1.67 (1.303) | -1.44 (1.000) | -0.80 (0.687) | -0.95 (0.891) | -0.97 (1.361)
  Week 96: number analyzed (Participants) | 26 | 27 | 24 | 26 | 14 | 13
  Week 96 | -1.55 (1.334) | -1.58 (1.325) | -1.43 (1.092) | -0.84 (0.710) | -1.21 (1.104) | -1.07 (1.357)

29. Secondary Outcome: Change From Baseline in HBV DNA Levels
Description: Change from baseline in HBV DNA levels were reported.
Time Frame: Baseline, Weeks 12, 24, 48, 60, 72, 96
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | Arm 1: JNJ-73763989 100 mg + JNJ-56136379 250 mg + NA | Arm 2: JNJ-73763989 200 mg + Placebo + NA | Arm 3: JNJ-73763989 100 mg + Placebo + NA | Arm 4: JNJ-73763989 40 mg + Placebo + NA | Arm 5: Placebo + JNJ-56136379 250 mg + NA | Arm 6: Placebo + Placebo + NA
Number analyzed (Participants) | 33 | 35 | 33 | 33 | 18 | 16
log10 IU/mL
  Baseline | 5.97 (1.989) | 6.64 (1.972) | 6.34 (1.778) | 6.10 (1.916) | 6.48 (2.008) | 6.39 (1.922)
  Week 12: number analyzed (Participants) | 33 | 34 | 33 | 31 | 16 | 16
  Week 12 | -4.13 (1.267) | -3.90 (1.221) | -3.83 (1.079) | -3.72 (1.008) | -4.28 (1.052) | -3.64 (1.365)
  Week 24: number analyzed (Participants) | 32 | 33 | 32 | 31 | 16 | 16
  Week 24 | -4.59 (1.532) | -5.03 (1.441) | -4.68 (1.199) | -4.53 (1.273) | -5.08 (1.566) | -4.34 (1.457)
  Week 48: number analyzed (Participants) | 30 | 32 | 32 | 30 | 15 | 16
  Week 48 | -4.85 (1.896) | -5.28 (1.663) | -5.18 (1.669) | -4.86 (1.605) | -5.71 (1.578) | -4.68 (1.970)
  Week 60: number analyzed (Participants) | 31 | 32 | 28 | 31 | 17 | 16
  Week 60 | -4.85 (1.910) | -5.39 (1.673) | -5.27 (1.759) | -4.95 (1.602) | -5.40 (1.808) | -4.67 (2.028)
  Week 72: number analyzed (Participants) | 30 | 31 | 29 | 31 | 17 | 16
  Week 72 | -4.97 (1.912) | -5.40 (1.849) | -5.25 (1.727) | -5.04 (1.606) | -5.49 (1.845) | -4.81 (1.903)
  Week 96: number analyzed (Participants) | 31 | 30 | 29 | 28 | 17 | 16
  Week 96 | -4.96 (2.010) | -5.45 (1.948) | -5.18 (2.004) | -5.06 (1.693) | -5.63 (1.827) | -4.95 (1.963)

30. Secondary Outcome: Time to Achieve HBsAg Seroclearance
Description: Time to HBsAg seroclearance (defined as HBsAg level <LLOQ [0.05 IU/mL]) was defined as the number of days between the date of first study treatment intake and the date of the first occurrence of HBsAg seroclearance.
Time Frame: Baseline (Day 1) up to Week 96
Population: mITT set: participants who were randomized in study and received at least one dose of study treatment excluding those participants impacted by pandemic because of COVID-19 or similar pandemics related reasons, withdrew prematurely from study prior to Week 44. N (number of participants analyzed): participants who achieved seroclearance and were available for the analysis and '0' in the number of participants analyzed field signifies none of the participant achieved seroclearance.
Measure: Median (90% Confidence Interval); unit: Weeks
Arm/Group | Arm 1: JNJ-73763989 100 mg + JNJ-56136379 250 mg + NA | Arm 2: JNJ-73763989 200 mg + Placebo + NA | Arm 3: JNJ-73763989 100 mg + Placebo + NA | Arm 4: JNJ-73763989 40 mg + Placebo + NA | Arm 5: Placebo + JNJ-56136379 250 mg + NA | Arm 6: Placebo + Placebo + NA
Number analyzed (Participants) | 0 | 5 | 3 | 0 | 0 | 1
Weeks |  | NA [NA to NA] — Here "NA" signifies that median and 90% confidence interval (CI) could not be calculated due to insufficient number of participants with events. | NA [NA to NA] — Here "NA" signifies that median and 90% CI could not be calculated due to insufficient number of participants with events. |  |  | NA [NA to NA] — Here "NA" signifies that median and 90% CI could not be calculated due to insufficient number of participants with events.

31. Secondary Outcome: Time to Achieve HBeAg Seroclearance
Description: Time to HBeAg seroclearance (defined as HBeAg level <LLOQ [0.11 IU/mL]) was defined as the number of days between the date of first study treatment intake and the date of the first occurrence of HBeAg seroclearance.
Time Frame: Baseline (Day 1) up to Week 96
Population: mITT analysis set: all participants who were randomized in study and received at least one dose of study treatment excluding those participants impacted by pandemic: those participants who, because of COVID-19 or similar pandemics related reasons, withdrew prematurely from study prior to Week 44. Here, 'Here, 'N' (number of participants analyzed) signifies HBeAg positive participants who achieved seroclearance and were available for the analysis
Measure: Median (90% Confidence Interval); unit: Weeks
Arm/Group | Arm 1: JNJ-73763989 100 mg + JNJ-56136379 250 mg + NA | Arm 2: JNJ-73763989 200 mg + Placebo + NA | Arm 3: JNJ-73763989 100 mg + Placebo + NA | Arm 4: JNJ-73763989 40 mg + Placebo + NA | Arm 5: Placebo + JNJ-56136379 250 mg + NA | Arm 6: Placebo + Placebo + NA
Number analyzed (Participants) | 6 | 5 | 7 | 3 | 4 | 2
Weeks | NA [NA to NA] — Here "NA" signifies that median, lower and upper limit of 90% confidence interval (CI) could not be calculated due to insufficient number of participants with events. | NA [NA to NA] — Here "NA" signifies that median, lower and upper limit of 90% CI could not be calculated due to insufficient number of participants with events. | NA [NA to NA] — Here "NA" signifies that median, lower and upper limit of 90% CI could not be calculated due to insufficient number of participants with events. | NA [NA to NA] — Here "NA" signifies that median, lower and upper limit of 90% CI could not be calculated due to insufficient number of participants with events. | NA [NA to NA] — Here "NA" signifies that median, lower and upper limit of 90% CI could not be calculated due to insufficient number of participants with events. | NA [NA to NA] — Here "NA" signifies that median, lower and upper limit of 90% CI could not be calculated due to insufficient number of participants with events.

32. Secondary Outcome: Percentage of Participants With HBsAg Levels <100 IU/mL
Description: Percentage of participants with HBsAg levels <100 IU/mL was reported.
Time Frame: Baseline, Weeks 12, 24, 48, 60, 72, 96
Population: as for outcome 19
Measure: Number; unit: Percentage of participants
Arm/Group | Arm 1: JNJ-73763989 100 mg + JNJ-56136379 250 mg + NA | Arm 2: JNJ-73763989 200 mg + Placebo + NA | Arm 3: JNJ-73763989 100 mg + Placebo + NA | Arm 4: JNJ-73763989 40 mg + Placebo + NA | Arm 5: Placebo + JNJ-56136379 250 mg + NA | Arm 6: Placebo + Placebo + NA
Number analyzed (Participants) | 94 | 94 | 92 | 91 | 48 | 45
Percentage of participants
  Baseline | 0 | 1.1 | 1.1 | 0 | 0 | 0
  Week 12: number analyzed (Participants) | 92 | 92 | 86 | 88 | 45 | 45
  Week 12 | 19.6 | 33.7 | 30.2 | 15.9 | 0 | 0
  Week 24: number analyzed (Participants) | 91 | 92 | 88 | 88 | 45 | 44
  Week 24 | 42.9 | 65.2 | 59.1 | 25.0 | 0 | 0
  Week 48: number analyzed (Participants) | 87 | 91 | 88 | 86 | 45 | 44
  Week 48 | 57.5 | 74.7 | 69.3 | 36.0 | 0 | 2.3
  Week 60: number analyzed (Participants) | 87 | 85 | 84 | 83 | 46 | 45
  Week 60 | 54.0 | 61.2 | 56.0 | 22.9 | 0 | 2.2
  Week 72: number analyzed (Participants) | 85 | 83 | 82 | 84 | 46 | 45
  Week 72 | 43.5 | 47.0 | 37.8 | 14.3 | 0 | 2.2
  Week 96: number analyzed (Participants) | 89 | 82 | 85 | 82 | 44 | 45
  Week 96 | 21.3 | 35.4 | 28.2 | 9.8 | 0 | 2.2

33. Secondary Outcome: Percentage of Participants With HBsAg Levels >1 log10 IU/mL Reduction From Baseline
Description: Percentage of participants with HBsAg levels >1 log10 IU/mL reduction from baseline was reported.
Time Frame: Weeks 12, 24, 48, 60, 72, 96
Population: as for outcome 25
Measure: Number; unit: Percentage of partcipants
Arm/Group | Arm 1: JNJ-73763989 100 mg + JNJ-56136379 250 mg + NA | Arm 2: JNJ-73763989 200 mg + Placebo + NA | Arm 3: JNJ-73763989 100 mg + Placebo + NA | Arm 4: JNJ-73763989 40 mg + Placebo + NA | Arm 5: Placebo + JNJ-56136379 250 mg + NA | Arm 6: Placebo + Placebo + NA
Number analyzed (Participants) | 92 | 92 | 88 | 88 | 46 | 45
Percentage of partcipants
  Week 12: number analyzed (Participants) | 92 | 92 | 86 | 88 | 45 | 45
  Week 12 | 40.2 | 72.8 | 60.5 | 27.3 | 2.2 | 0
  Week 24: number analyzed (Participants) | 91 | 92 | 88 | 88 | 45 | 44
  Week 24 | 84.6 | 97.8 | 93.2 | 71.6 | 4.4 | 4.5
  Week 48: number analyzed (Participants) | 87 | 91 | 88 | 86 | 45 | 44
  Week 48 | 93.1 | 97.8 | 97.7 | 82.6 | 4.4 | 4.5
  Week 60: number analyzed (Participants) | 87 | 85 | 84 | 83 | 46 | 45
  Week 60 | 86.2 | 94.1 | 90.5 | 67.5 | 4.3 | 4.4
  Week 72: number analyzed (Participants) | 85 | 83 | 82 | 84 | 46 | 45
  Week 72 | 71.8 | 84.4 | 73.2 | 46.6 | 4.3 | 6.7
  Week 96: number analyzed (Participants) | 89 | 82 | 85 | 82 | 44 | 45
  Week 96 | 41.6 | 63.4 | 49.4 | 20.7 | 4.5 | 4.4

34. Secondary Outcome: Percentage of HBeAg-positive Participants With HBeAg Levels <LLOQ
Description: Percentage of HBeAg-positive participants with HBeAg levels <LLOQ were reported.
Time Frame: Weeks 12, 24, 48, 60, 72, 96
Population: as for outcome 25
Measure: Number; unit: Percentage of participants
Arm/Group | Arm 1: JNJ-73763989 100 mg + JNJ-56136379 250 mg + NA | Arm 2: JNJ-73763989 200 mg + Placebo + NA | Arm 3: JNJ-73763989 100 mg + Placebo + NA | Arm 4: JNJ-73763989 40 mg + Placebo + NA | Arm 5: Placebo + JNJ-56136379 250 mg + NA | Arm 6: Placebo + Placebo + NA
Number analyzed (Participants) | 27 | 29 | 25 | 30 | 15 | 13
Percentage of participants
  Week 12: number analyzed (Participants) | 27 | 27 | 23 | 29 | 13 | 10
  Week 12 | 7.4 | 3.7 | 17.4 | 6.9 | 7.7 | 0
  Week 24: number analyzed (Participants) | 27 | 29 | 25 | 30 | 13 | 13
  Week 24 | 7.4 | 3.4 | 16.0 | 6.7 | 7.7 | 0
  Week 48: number analyzed (Participants) | 26 | 28 | 24 | 27 | 14 | 13
  Week 48 | 19.2 | 7.1 | 20.8 | 11.1 | 7.1 | 15.4
  Week 60: number analyzed (Participants) | 25 | 27 | 24 | 27 | 15 | 12
  Week 60 | 12.0 | 11.1 | 16.7 | 7.4 | 6.7 | 16.7
  Week 72: number analyzed (Participants) | 25 | 27 | 23 | 28 | 15 | 13
  Week 72 | 8.0 | 11.1 | 21.7 | 10.7 | 6.7 | 15.4
  Week 96: number analyzed (Participants) | 26 | 27 | 24 | 26 | 14 | 13
  Week 96 | 15.4 | 14.8 | 20.8 | 11.5 | 21.4 | 15.4

35. Secondary Outcome: Percentage of HBeAg-positive Participants With HBeAg Levels >1 log10 IU/mL
Description: Percentage of HBeAg-positive partcipants with HBeAg levels >1 log10 IU/mL were reported.
Time Frame: Weeks 12, 24, 48, 60, 72, 96
Population: mITT population. Here, 'N' (number of participants analyzed) signifies HBeAg + participants who were evaluable for this outcome measure and 'n' (number analyzed) represents participants evaluable at the specified timepoint.
Measure: Number; unit: Percentage of participants
Arm/Group | Arm 1: JNJ-73763989 100 mg + JNJ-56136379 250 mg + NA | Arm 2: JNJ-73763989 200 mg + Placebo + NA | Arm 3: JNJ-73763989 100 mg + Placebo + NA | Arm 4: JNJ-73763989 40 mg + Placebo + NA | Arm 5: Placebo + JNJ-56136379 250 mg + NA | Arm 6: Placebo + Placebo + NA
Number analyzed (Participants) | 27 | 29 | 25 | 30 | 15 | 13
Percentage of participants
  Week 12: number analyzed (Participants) | 27 | 27 | 23 | 29 | 13 | 10
  Week 12 | 33.3 | 33.3 | 39.1 | 3.4 | 23.1 | 10.0
  Week 24: number analyzed (Participants) | 27 | 29 | 25 | 30 | 13 | 13
  Week 24 | 44.4 | 48.3 | 60.0 | 10.0 | 30.8 | 23.1
  Week 48: number analyzed (Participants) | 26 | 28 | 24 | 27 | 14 | 13
  Week 48 | 50.0 | 53.6 | 66.7 | 25.9 | 35.7 | 30.8
  Week 60: number analyzed (Participants) | 25 | 27 | 24 | 27 | 15 | 12
  Week 60 | 52.0 | 63.3 | 62.5 | 37.0 | 40.0 | 33.3
  Week 72: number analyzed (Participants) | 25 | 27 | 23 | 28 | 15 | 13
  Week 72 | 56.0 | 59.3 | 65.2 | 35.7 | 40.0 | 30.8
  Week 96: number analyzed (Participants) | 26 | 27 | 24 | 26 | 14 | 13
  Week 96 | 53.8 | 59.3 | 58.3 | 42.3 | 42.9 | 30.8

36. Secondary Outcome: Percentage of Participants With HBV DNA Levels <LLOQ
Description: Percentage of participants with HBV DNA levels <LLOQ (20 IU/mL) were reported.
Time Frame: Baseline, Weeks 12, 24, 48, 60, 72, 96
Population: as for outcome 19
Measure: Number; unit: Percentage of participants
Arm/Group | Arm 1: JNJ-73763989 100 mg + JNJ-56136379 250 mg + NA | Arm 2: JNJ-73763989 200 mg + Placebo + NA | Arm 3: JNJ-73763989 100 mg + Placebo + NA | Arm 4: JNJ-73763989 40 mg + Placebo + NA | Arm 5: Placebo + JNJ-56136379 250 mg + NA | Arm 6: Placebo + Placebo + NA
Number analyzed (Participants) | 94 | 94 | 92 | 91 | 48 | 45
Percentage of participants
  Baseline | 64.4 | 60.4 | 63.7 | 60.9 | 60.6 | 63.8
  Week 12: number analyzed (Participants) | 92 | 92 | 86 | 88 | 45 | 45
  Week 12 | 78.3 | 71.7 | 76.7 | 70.5 | 73.3 | 75.6
  Week 24: number analyzed (Participants) | 91 | 92 | 88 | 88 | 45 | 44
  Week 24 | 84.6 | 80.4 | 81.8 | 83.0 | 80.0 | 77.3
  Week 48: number analyzed (Participants) | 88 | 91 | 88 | 87 | 45 | 45
  Week 48 | 92.0 | 85.7 | 86.4 | 90.8 | 95.6 | 93.3
  Week 60: number analyzed (Participants) | 88 | 85 | 83 | 85 | 46 | 45
  Week 60 | 88.6 | 85.9 | 79.5 | 85.9 | 93.5 | 93.3
  Week 72: number analyzed (Participants) | 86 | 85 | 83 | 84 | 46 | 45
  Week 72 | 89.5 | 81.2 | 81.9 | 86.9 | 95.7 | 91.1
  Week 96: number analyzed (Participants) | 89 | 82 | 85 | 80 | 44 | 45
  Week 96 | 94.4 | 75.6 | 80.0 | 87.5 | 95.5 | 93.3

37. Secondary Outcome: Mean Change From Baseline in ALT at EOT (Week 48) in Participants With Elevated ALT at Baseline
Description: Mean change from baseline in ALT at EOT (Week 48) in participants with elevated ALT at baseline were reported.
Time Frame: Baseline and Week 48
Population: mITT analysis set: all participants who were randomized in study and received at least one dose of study treatment excluding those participants impacted by pandemic: those participants who, because of COVID-19 or similar pandemics related reasons, withdrew prematurely from study prior to Week 44. Here, 'N' (number of participants analyzed) signifies participants with ALT elevation at baseline who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Units per liter (U/L)
Arm/Group | Arm 1: JNJ-73763989 100 mg + JNJ-56136379 250 mg + NA | Arm 2: JNJ-73763989 200 mg + Placebo + NA | Arm 3: JNJ-73763989 100 mg + Placebo + NA | Arm 4: JNJ-73763989 40 mg + Placebo + NA | Arm 5: Placebo + JNJ-56136379 250 mg + NA | Arm 6: Placebo + Placebo + NA
Number analyzed (Participants) | 35 | 32 | 37 | 34 | 19 | 18
Units per liter (U/L) | -72.77 (106.851) [lower limit 106.851] | -65.47 (110.213) [lower limit 110.213] | -37.51 (63.468) [lower limit 63.468] | -42.53 (41.767) [lower limit 41.767] | -17.68 (272.44) [lower limit 272.44] | -49.28 (85.374) [lower limit 85.374]

38. Secondary Outcome: Percentage of Participants With ALT Normalization
Description: Percentage of participants with ALT normalization was reported. A participant with ALT elevation at baseline was considered to achieve ALT normalization if his/her ALT value was <ULN at any given postbaseline analysis time point. A participant was defined as on treatment failure if he/she never met the criteria for stopping NA treatment during the study. A participant was defined as off-treatment failure if he/she required NA re-treatment after stopping all study interventions.
Time Frame: Baseline, Weeks 12, 24, 48, 60, 72, 96
Population: as for outcome 25
Measure: Number; unit: Percentage of participants
Arm/Group | Arm 1: JNJ-73763989 100 mg + JNJ-56136379 250 mg + NA | Arm 2: JNJ-73763989 200 mg + Placebo + NA | Arm 3: JNJ-73763989 100 mg + Placebo + NA | Arm 4: JNJ-73763989 40 mg + Placebo + NA | Arm 5: Placebo + JNJ-56136379 250 mg + NA | Arm 6: Placebo + Placebo + NA
Number analyzed (Participants) | 36 | 32 | 37 | 34 | 19 | 18
Percentage of participants
  Baseline | 0 | 0 | 0 | 0 | 0 | 0
  Week 12 On-treatment: number analyzed (Participants) | 35 | 31 | 36 | 31 | 16 | 17
  Week 12 On-treatment | 54.3 | 41.9 | 58.3 | 64.5 | 56.3 | 47.1
  Week 24 On-treatment: number analyzed (Participants) | 34 | 30 | 36 | 33 | 17 | 18
  Week 24 On-treatment | 61.8 | 43.3 | 69.4 | 78.8 | 76.5 | 55.6
  Week 48 On-treatment: number analyzed (Participants) | 33 | 30 | 35 | 31 | 16 | 17
  Week 48 On-treatment | 60.6 | 46.7 | 65.7 | 83.9 | 87.5 | 58.8
  Week 60 On-treatment: number analyzed (Participants) | 33 | 28 | 33 | 33 | 18 | 18
  Week 60 On-treatment | 0 | 3.6 | 12.1 | 0 | 0 | 5.6
  Week 72 On-treatment: number analyzed (Participants) | 32 | 28 | 33 | 33 | 18 | 18
  Week 72 On-treatment | 0 | 3.6 | 12.1 | 0 | 0 | 5.6
  Week 96 On-treatment: number analyzed (Participants) | 33 | 26 | 34 | 30 | 18 | 18
  Week 96 On-treatment | 21.2 | 11.5 | 35.3 | 10.0 | 16.7 | 11.1
  Week 60 Off-treatment: number analyzed (Participants) | 33 | 28 | 33 | 33 | 18 | 18
  Week 60 Off-treatment | 0 | 3.6 | 12.1 | 0 | 0 | 5.6
  Week 72 Off-treatment: number analyzed (Participants) | 32 | 28 | 33 | 33 | 18 | 18
  Week 72 Off-treatment | 0 | 3.6 | 12.1 | 0 | 0 | 5.6
  Week 96 Off-treatment: number analyzed (Participants) | 33 | 26 | 34 | 30 | 18 | 18
  Week 96 Off-treatment | 21.2 | 11.5 | 35.3 | 10.0 | 16.7 | 11.1

39. Secondary Outcome: Percentage of Participants With Virologic Breakthrough
Description: Virologic breakthrough was defined as having a confirmed on-treatment HBV DNA increase by >1 log10 from nadir (that is, lowest value during treatment) or a confirmed HBV DNA level >200 IU/mL in participants who had on-treatment HBV DNA level below the LLOQ (20 IU/mL). On-treatment was defined as the time period in which the participant received any of the study intervention.
Time Frame: Baseline (Day 1) up to Week 48
Population: mITT analysis set: all participants who were randomized in study and received at least one dose of study treatment excluding those participants impacted by pandemic: those participants who, because of COVID-19 or similar pandemics related reasons, withdrew prematurely from study prior to Week 44.
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm 1: JNJ-73763989 100 mg + JNJ-56136379 250 mg + NA | Arm 2: JNJ-73763989 200 mg + Placebo + NA | Arm 3: JNJ-73763989 100 mg + Placebo + NA | Arm 4: JNJ-73763989 40 mg + Placebo + NA | Arm 5: Placebo + JNJ-56136379 250 mg + NA | Arm 6: Placebo + Placebo + NA
Number analyzed (Participants) | 94 | 94 | 92 | 91 | 48 | 45
Percentage of participants | 2.1 (0.38) [0.38 to 6.55] | 2.1 (0.38) [0.38 to 6.55] | 2.2 (0.39) [0.39 to 6.69] | 2.2 (0.39) [0.39 to 6.76] | 0.0 (0.00) [0.00 to 6.05] | 2.2 (0.11) [0.11 to 10.11]

40. Secondary Outcome: Percentage of Participants With Undetectable HBV DNA Levels After Re-start of NA Treatment During Follow-up
Description: Percentage of participants with undetectable HBV DNA levels after re-start of NA treatment during follow-up was reported.
Time Frame: Week 48 up to Week 96
Population: as for outcome 39
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm 1: JNJ-73763989 100 mg + JNJ-56136379 250 mg + NA | Arm 2: JNJ-73763989 200 mg + Placebo + NA | Arm 3: JNJ-73763989 100 mg + Placebo + NA | Arm 4: JNJ-73763989 40 mg + Placebo + NA | Arm 5: Placebo + JNJ-56136379 250 mg + NA | Arm 6: Placebo + Placebo + NA
Number analyzed (Participants) | 94 | 94 | 92 | 91 | 48 | 45
Percentage of participants | 1.1 (0.05) [0.05 to 4.95] | 1.1 (0.05) [0.05 to 4.95] | 1.1 (0.06) [0.06 to 5.05] | 0.0 (0.00) [0.00 to 3.24] | 0.0 (0.00) [0.00 to 6.05] | 0.0 (0.00) [0.00 to 6.44]

ADVERSE EVENTS:
Time Frame: Double blind (DB) phase: Baseline (Day 1) up to Week 48, Follow up (FU) phase: Week 48 up to Week 96; Extended Follow-up Phase: Extended follow up Week 1 to extended follow-up Week 48
Description: Safety analysis set included all participants who received at least one dose of any of the study treatments. At risk = 0 signifies that none of the participant in that arm entered the respective follow up phase.
Groups:
- Arm 1: DB Phase: JNJ-73763989 100 mg + JNJ-56136379 250 mg + NA: Participants received JNJ-73763989 100 milligrams (mg) as subcutaneous (SC) injection once every 4 weeks along with JNJ-56136379 250 mg as oral tablet once daily and Nucleos(t)ide Analog (NA) (either entecavir [ETV] monohydrate 0.5 mg, tenofovir disoproxil fumarate [TDF] 300 mg, or tenofovir alafenamide [TAF] 25 mg) tablet orally once daily up to 48 weeks.
- Arm 2: DB Phase: JNJ-73763989 200 mg + Placebo + NA: Participants with CHB received JNJ-73763989 200 mg as SC injection once every 4 weeks along with placebo matching to JNJ-56136379 tablet orally once daily and NA (either ETV 0.5 mg, TDF 300 mg, or TAF 25 mg) tablet orally once daily up to 48 weeks.
- Arm 3: DB Phase: JNJ-73763989 (100 mg) + Placebo + NA: Participants received JNJ-73763989 100 mg as SC injection once every 4 weeks along with placebo matching to JNJ-56136379 tablet orally and NA (either ETV 0.5 mg, TDF 300 mg, or TAF 25 mg) tablets orally once daily up to 48 weeks.
- Arm 4: DB Phase: JNJ-73763989 (40 mg) + Placebo + NA: Participants received JNJ-73763989 40 mg as SC injection once every 4 weeks along with placebo matching to JNJ-56136379 tablet orally and NA (either ETV 0.5 mg, TDF 300 mg, or TAF 25 mg) tablet orally once daily up to 48 weeks.
- Arm 5: DB Phase: Placebo + JNJ-56136379 250 mg + NA: Participants received placebo matching to JNJ-73763989 as SC injection and a fixed dose of JNJ-56136379 250 mg oral tablet once daily along with NA (either ETV 0.5 mg, TDF 300 mg, or TAF 25 mg) tablet orally once daily up to 48 weeks.
- Arm 6: DB Phase: Placebo + Placebo + NA: Participants received placebo matching to JNJ-73763989 as SC injection and placebo matching to JNJ-56136379 tablet orally along with NA (either ETV 0.5 mg, TDF 300 mg, or TAF 25 mg) tablet orally once daily up to 48 weeks.
Arm/Group | Arm 1: DB Phase: JNJ-73763989 100 mg + JNJ-56136379 250 mg + NA | Arm 2: DB Phase: JNJ-73763989 200 mg + Placebo + NA | Arm 3: DB Phase: JNJ-73763989 (100 mg) + Placebo + NA | Arm 4: DB Phase: JNJ-73763989 (40 mg) + Placebo + NA | Arm 5: DB Phase: Placebo + JNJ-56136379 250 mg + NA | Arm 6: DB Phase: Placebo + Placebo + NA | Arm 1: Follow up Phase 1: JNJ-73763989 (100 mg) + JNJ-56136379 (250 mg) + NA | Arm 2: Follow up Phase 1: JNJ-73763989 (200mg) + Placebo + NA | Arm 3: Follow up Phase 1: JNJ-73763989 (100 mg) + Placebo + NA | Arm 4: Follow up Phase 1: JNJ-73763989 (40 mg) + Placebo + NA | Arm 5: Follow up Phase 1: Placebo + JNJ-56136379 250 mg + NA | Arm 6 :Follow up Phase 1: Placebo + Placebo + NA | Arm 1: Follow up Phase 2: JNJ-73763989 (100 mg) + JNJ-56136379 (250 mg) + NA | Arm 2: Follow up Phase 2: JNJ-73763989 (200mg) + Placebo + NA | Arm 3: Follow up Phase 2: JNJ-73763989 (100 mg) + Placebo + NA | Arm 4: Follow up Phase 2: JNJ-73763989 (40 mg) + Placebo + NA | Arm 5: Follow up Phase 2: Placebo + JNJ-56136379 250 mg + NA | Arm 6: Follow up Phase 2: Placebo + Placebo + NA | Arm 1: Follow up Phase 3: JNJ-73763989 (100 mg) + JNJ-56136379 (250 mg) + NA | Arm 2: Follow up Period 3: JNJ-73763989 (200mg) + Placebo + NA | Arm 3: Follow up Phase 3: JNJ-73763989 (100 mg) + Placebo + NA | Arm 4: Follow up Phase 3: JNJ-73763989 (40 mg) + Placebo + NA | Arm 5: Follow up Phase 3: Placebo + JNJ-56136379 250 mg + NA | Arm 6: Follow up Phase 3: Placebo + Placebo + NA | Arm 1: Extended Follow up: JNJ-73763989 (100 mg) + JNJ-56136379 (250 mg) + NA | Arm 2: Extended Follow Up: JNJ-73763989 (200 mg) + Placebo + NA | Arm 3: Extended Follow up: JNJ-73763989 (100 mg) + Placebo + NA | Arm 4: Extended Follow Up: JNJ-73763989 (40 mg) + Placebo + NA | Arm 5: Extended Follow Up: Placebo + JNJ-56136379 250 mg + NA | Arm 6: Extended Follow Up: Placebo + Placebo + NA
All-Cause Mortality (participants affected / at risk) | 0/95 | 0/96 | 0/93 | 0/93 | 0/48 | 0/45 | 0/81 | 0/70 | 0/71 | 0/85 | 0/47 | 0/44 | 0/8 | 0/17 | 0/15 | 0/5 | 0/0 | 0/1 | 0/3 | 0/8 | 0/5 | 0/0 | 0/0 | 0/0 | 0/3 | 0/7 | 0/5 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 2/95 | 3/96 | 2/93 | 1/93 | 2/48 | 0/45 | 1/81 | 5/70 | 3/71 | 1/85 | 1/47 | 0/44 | 1/8 | 0/17 | 0/15 | 0/5 | 0/0 | 0/1 | 1/3 | 0/8 | 0/5 | 0/0 | 0/0 | 0/0 | 0/3 | 1/7 | 2/5 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 66/95 | 59/96 | 59/93 | 60/93 | 41/48 | 30/45 | 28/81 | 28/70 | 35/71 | 32/85 | 26/47 | 14/44 | 3/8 | 5/17 | 9/15 | 3/5 | 0/0 | 0/1 | 1/3 | 3/8 | 1/5 | 0/0 | 0/0 | 0/0 | 2/3 | 5/7 | 5/5 | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: DB Phase: JNJ-73763989 100 mg + JNJ-56136379 250 mg + NA (N=95) | Arm 2: DB Phase: JNJ-73763989 200 mg + Placebo + NA (N=96) | Arm 3: DB Phase: JNJ-73763989 (100 mg) + Placebo + NA (N=93) | Arm 4: DB Phase: JNJ-73763989 (40 mg) + Placebo + NA (N=93) | Arm 5: DB Phase: Placebo + JNJ-56136379 250 mg + NA (N=48) | Arm 6: DB Phase: Placebo + Placebo + NA (N=45) | Arm 1: Follow up Phase 1: JNJ-73763989 (100 mg) + JNJ-56136379 (250 mg) + NA (N=81) | Arm 2: Follow up Phase 1: JNJ-73763989 (200mg) + Placebo + NA (N=70) | Arm 3: Follow up Phase 1: JNJ-73763989 (100 mg) + Placebo + NA (N=71) | Arm 4: Follow up Phase 1: JNJ-73763989 (40 mg) + Placebo + NA (N=85) | Arm 5: Follow up Phase 1: Placebo + JNJ-56136379 250 mg + NA (N=47) | Arm 6 :Follow up Phase 1: Placebo + Placebo + NA (N=44) | Arm 1: Follow up Phase 2: JNJ-73763989 (100 mg) + JNJ-56136379 (250 mg) + NA (N=8) | Arm 2: Follow up Phase 2: JNJ-73763989 (200mg) + Placebo + NA (N=17) | Arm 3: Follow up Phase 2: JNJ-73763989 (100 mg) + Placebo + NA (N=15) | Arm 4: Follow up Phase 2: JNJ-73763989 (40 mg) + Placebo + NA (N=5) | Arm 5: Follow up Phase 2: Placebo + JNJ-56136379 250 mg + NA (N=0) | Arm 6: Follow up Phase 2: Placebo + Placebo + NA (N=1) | Arm 1: Follow up Phase 3: JNJ-73763989 (100 mg) + JNJ-56136379 (250 mg) + NA (N=3) | Arm 2: Follow up Period 3: JNJ-73763989 (200mg) + Placebo + NA (N=8) | Arm 3: Follow up Phase 3: JNJ-73763989 (100 mg) + Placebo + NA (N=5) | Arm 4: Follow up Phase 3: JNJ-73763989 (40 mg) + Placebo + NA (N=0) | Arm 5: Follow up Phase 3: Placebo + JNJ-56136379 250 mg + NA (N=0) | Arm 6: Follow up Phase 3: Placebo + Placebo + NA (N=0) | Arm 1: Extended Follow up: JNJ-73763989 (100 mg) + JNJ-56136379 (250 mg) + NA (N=3) | Arm 2: Extended Follow Up: JNJ-73763989 (200 mg) + Placebo + NA (N=7) | Arm 3: Extended Follow up: JNJ-73763989 (100 mg) + Placebo + NA (N=5) | Arm 4: Extended Follow Up: JNJ-73763989 (40 mg) + Placebo + NA (N=0) | Arm 5: Extended Follow Up: Placebo + JNJ-56136379 250 mg + NA (N=0) | Arm 6: Extended Follow Up: Placebo + Placebo + NA (N=0)
Coronary Artery Disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Retinal Detachment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Gastric Polyps (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 1 | NA | NA | NA
Gastric Ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Melaena (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Cholecystitis Chronic (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 1 | 0 | NA | NA | NA
Gallbladder Cholesterolosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 1 | 0 | NA | NA | NA
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 1 | NA | NA | NA
Covid-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Covid-19 Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Pneumocystis Jirovecii Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Urinary Tract Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Fracture Displacement (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Ligament Rupture (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Multiple Injuries (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Tibia Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Alanine Aminotransferase Increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Aspartate Aminotransferase Increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Hepatocellular Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | NA | 0 | 1 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Myoclonus (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Renal Colic (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Urinary Incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: DB Phase: JNJ-73763989 100 mg + JNJ-56136379 250 mg + NA (N=95) | Arm 2: DB Phase: JNJ-73763989 200 mg + Placebo + NA (N=96) | Arm 3: DB Phase: JNJ-73763989 (100 mg) + Placebo + NA (N=93) | Arm 4: DB Phase: JNJ-73763989 (40 mg) + Placebo + NA (N=93) | Arm 5: DB Phase: Placebo + JNJ-56136379 250 mg + NA (N=48) | Arm 6: DB Phase: Placebo + Placebo + NA (N=45) | Arm 1: Follow up Phase 1: JNJ-73763989 (100 mg) + JNJ-56136379 (250 mg) + NA (N=81) | Arm 2: Follow up Phase 1: JNJ-73763989 (200mg) + Placebo + NA (N=70) | Arm 3: Follow up Phase 1: JNJ-73763989 (100 mg) + Placebo + NA (N=71) | Arm 4: Follow up Phase 1: JNJ-73763989 (40 mg) + Placebo + NA (N=85) | Arm 5: Follow up Phase 1: Placebo + JNJ-56136379 250 mg + NA (N=47) | Arm 6 :Follow up Phase 1: Placebo + Placebo + NA (N=44) | Arm 1: Follow up Phase 2: JNJ-73763989 (100 mg) + JNJ-56136379 (250 mg) + NA (N=8) | Arm 2: Follow up Phase 2: JNJ-73763989 (200mg) + Placebo + NA (N=17) | Arm 3: Follow up Phase 2: JNJ-73763989 (100 mg) + Placebo + NA (N=15) | Arm 4: Follow up Phase 2: JNJ-73763989 (40 mg) + Placebo + NA (N=5) | Arm 5: Follow up Phase 2: Placebo + JNJ-56136379 250 mg + NA (N=0) | Arm 6: Follow up Phase 2: Placebo + Placebo + NA (N=1) | Arm 1: Follow up Phase 3: JNJ-73763989 (100 mg) + JNJ-56136379 (250 mg) + NA (N=3) | Arm 2: Follow up Period 3: JNJ-73763989 (200mg) + Placebo + NA (N=8) | Arm 3: Follow up Phase 3: JNJ-73763989 (100 mg) + Placebo + NA (N=5) | Arm 4: Follow up Phase 3: JNJ-73763989 (40 mg) + Placebo + NA (N=0) | Arm 5: Follow up Phase 3: Placebo + JNJ-56136379 250 mg + NA (N=0) | Arm 6: Follow up Phase 3: Placebo + Placebo + NA (N=0) | Arm 1: Extended Follow up: JNJ-73763989 (100 mg) + JNJ-56136379 (250 mg) + NA (N=3) | Arm 2: Extended Follow Up: JNJ-73763989 (200 mg) + Placebo + NA (N=7) | Arm 3: Extended Follow up: JNJ-73763989 (100 mg) + Placebo + NA (N=5) | Arm 4: Extended Follow Up: JNJ-73763989 (40 mg) + Placebo + NA (N=0) | Arm 5: Extended Follow Up: Placebo + JNJ-56136379 250 mg + NA (N=0) | Arm 6: Extended Follow Up: Placebo + Placebo + NA (N=0)
Anaemia (Blood and lymphatic system disorders) | 2 | 2 | 3 | 3 | 1 | 3 | 1 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Atrioventricular Block First Degree (Cardiac disorders) | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Palpitations (Cardiac disorders) | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Supraventricular Extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Ear Pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Otosclerosis (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Thyroid Cyst (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 1 | NA | NA | NA
Blepharospasm (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Chorioretinal Scar (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Conjunctivitis Allergic (Eye disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Dry Eye (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Photophobia (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Photopsia (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Strabismus (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 1 | NA | NA | NA
Vision Blurred (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Abdominal Discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Abdominal Distension (Gastrointestinal disorders) | 1 | 2 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Abdominal Pain (Gastrointestinal disorders) | 1 | 0 | 5 | 4 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Abdominal Pain Lower (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Abdominal Pain Upper (Gastrointestinal disorders) | 3 | 3 | 2 | 2 | 1 | 2 | 0 | 2 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Abnormal Faeces (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Aphthous Ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Chronic Gastritis (Gastrointestinal disorders) | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Constipation (Gastrointestinal disorders) | 3 | 2 | 3 | 1 | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Dental Caries (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Diarrhoea (Gastrointestinal disorders) | 4 | 3 | 10 | 4 | 2 | 2 | 0 | 1 | 1 | 3 | 2 | 0 | 1 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Diarrhoea Haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Dry Mouth (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Dyspepsia (Gastrointestinal disorders) | 1 | 3 | 2 | 4 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 1 | NA | NA | NA
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Epigastric Discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Frequent Bowel Movements (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 1 | NA | NA | NA | 0 | 0 | 1 | NA | NA | NA
Gastrointestinal Erosion (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 1 | NA | NA | NA
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Gingival Swelling (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Glossitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Haemorrhoidal Haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Haemorrhoids (Gastrointestinal disorders) | 1 | 3 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 1 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Haemorrhoids Thrombosed (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Mouth Ulceration (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Nausea (Gastrointestinal disorders) | 4 | 7 | 6 | 6 | 6 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Tooth Disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Toothache (Gastrointestinal disorders) | 2 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Vomiting (Gastrointestinal disorders) | 1 | 2 | 2 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Asthenia (General disorders) | 2 | 5 | 5 | 2 | 4 | 4 | 1 | 2 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Chest Pain (General disorders) | 1 | 1 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Chills (General disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Fatigue (General disorders) | 7 | 2 | 3 | 5 | 6 | 3 | 1 | 1 | 1 | 2 | 1 | 0 | 0 | 0 | 1 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Feeling Hot (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Influenza Like Illness (General disorders) | 1 | 3 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Injection Site Bruising (General disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Injection Site Erythema (General disorders) | 2 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Injection Site Pain (General disorders) | 2 | 0 | 6 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Injection Site Reaction (General disorders) | 3 | 2 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Malaise (General disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | NA | 0 | 0 | 1 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Non-Cardiac Chest Pain (General disorders) | 0 | 4 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Oedema Peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 1 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Peripheral Swelling (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Pyrexia (General disorders) | 2 | 1 | 1 | 2 | 2 | 1 | 2 | 3 | 2 | 1 | 3 | 1 | 0 | 1 | 1 | 1 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 2 | 0 | NA | NA | NA
Thirst (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Vaccination Site Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Deficiency of Bile Secretion (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Hepatic Cyst (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Hepatic Steatosis (Hepatobiliary disorders) | 0 | 1 | 2 | 2 | 0 | 0 | 1 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 2 | NA | NA | NA
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Contrast Media Allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Seasonal Allergy (Immune system disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Campylobacter Colitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Conjunctivitis (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 1 | NA | NA | NA
Covid-19 (Infections and infestations) | 4 | 4 | 3 | 2 | 1 | 2 | 3 | 8 | 7 | 8 | 5 | 4 | 0 | 0 | 1 | 1 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 1 | 0 | 0 | NA | NA | NA
Ear Infection (Infections and infestations) | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Epididymitis (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Eyelid Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Fungal Infection (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Furuncle (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Gastroenteritis Viral (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Genital Herpes (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Helicobacter Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 1 | NA | NA | NA
Influenza (Infections and infestations) | 1 | 3 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 1 | NA | NA | NA
Localised Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 1 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Nasopharyngitis (Infections and infestations) | 6 | 4 | 8 | 5 | 3 | 1 | 3 | 1 | 3 | 3 | 1 | 0 | 0 | 0 | 1 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 1 | 0 | NA | NA | NA
Oral Candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Oral Herpes (Infections and infestations) | 0 | 2 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Periodontitis (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 1 | NA | NA | NA
Pharyngitis (Infections and infestations) | 2 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Pulpitis Dental (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Respiratory Tract Infection (Infections and infestations) | 2 | 3 | 0 | 2 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Respiratory Tract Infection Viral (Infections and infestations) | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Rhinitis (Infections and infestations) | 1 | 1 | 1 | 1 | 3 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Skin Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Tooth Abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Tooth Infection (Infections and infestations) | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Upper Respiratory Tract Infection (Infections and infestations) | 2 | 3 | 4 | 3 | 2 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 1 | NA | NA | NA
Urinary Tract Infection (Infections and infestations) | 1 | 2 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 1 | 0 | 0 | NA | NA | NA
Varicella (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Viral Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Viral Upper Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Vulvovaginal Candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Animal Bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Arthropod Bite (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Contusion (Injury, poisoning and procedural complications) | 0 | 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Foot Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Head Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Joint Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 1 | NA | NA | NA
Ligament Sprain (Injury, poisoning and procedural complications) | 2 | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Limb Injury (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Muscle Strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Skin Abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Tendon Rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Thermal Burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Traumatic Tooth Displacement (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Ulna Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Upper Limb Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Vaccination Complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 1 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Alanine Aminotransferase Increased (Investigations) | 5 | 3 | 1 | 1 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Amylase Increased (Investigations) | 1 | 1 | 1 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Aspartate Aminotransferase Increased (Investigations) | 2 | 2 | 0 | 2 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Beta 2 Microglobulin Increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Blood Bicarbonate Decreased (Investigations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Blood Cholesterol Increased (Investigations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Blood Creatine Phosphokinase Increased (Investigations) | 2 | 1 | 2 | 1 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Blood Pressure Increased (Investigations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Blood Uric Acid Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Coagulation Time Prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Creatinine Renal Clearance Decreased (Investigations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Glomerular Filtration Rate Decreased (Investigations) | 11 | 2 | 5 | 5 | 3 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Haemoglobin Decreased (Investigations) | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Lipase Increased (Investigations) | 1 | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Serum Ferritin Decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Transaminases Increased (Investigations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Vitamin D Decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Weight Decreased (Investigations) | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 1 | 0 | NA | NA | NA
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 1 | 0 | NA | NA | NA | 0 | 1 | 0 | NA | NA | NA
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 1 | 0 | NA | NA | NA
Vitamin D Deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 3 | 3 | 6 | 1 | 1 | 2 | 1 | 3 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Back Pain (Musculoskeletal and connective tissue disorders) | 5 | 5 | 6 | 6 | 2 | 1 | 1 | 1 | 4 | 3 | 3 | 0 | 1 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Joint Range of Motion Decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 4 | 4 | 4 | 3 | 2 | 2 | 2 | 2 | 0 | 1 | 1 | 1 | 0 | 2 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 1 | NA | NA | NA
Pain in Jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Spinal Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Spinal Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Adenoma Benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Dizziness (Nervous system disorders) | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Dizziness Postural (Nervous system disorders) | 1 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Dysgeusia (Nervous system disorders) | 1 | 1 | 2 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Facial Spasm (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Headache (Nervous system disorders) | 13 | 12 | 17 | 14 | 4 | 7 | 2 | 3 | 3 | 2 | 2 | 0 | 0 | 1 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 1 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Sciatica (Nervous system disorders) | 1 | 0 | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Somnolence (Nervous system disorders) | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Anxiety (Psychiatric disorders) | 1 | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Confusional State (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Depressed Mood (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Depression (Psychiatric disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Insomnia (Psychiatric disorders) | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Sleep Disorder (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Azotaemia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Calculus Urinary (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Dysuria (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Glycosuria (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Leukocyturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Renal Impairment (Renal and urinary disorders) | 3 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Renal Pain (Renal and urinary disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Atrophic Vulvovaginitis (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Cervical Dysplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Erectile Dysfunction (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Heavy Menstrual Bleeding (Reproductive system and breast disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Menstruation Irregular (Reproductive system and breast disorders) | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Pruritus Genital (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 1 | 0 | NA | NA | NA
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 5 | 3 | 3 | 2 | 3 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Cystic Lung Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 1 | NA | NA | NA
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Nasal Dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 3 | 0 | 3 | 1 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Pulmonary Mass (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 1 | NA | NA | NA
Respiratory Disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Alopecia (Skin and subcutaneous tissue disorders) | 5 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Dry Skin (Skin and subcutaneous tissue disorders) | 2 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Eczema Asteatotic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Hyperkeratosis Follicularis Et Parafollicularis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Hypertrichosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Nail Disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Photosensitivity Reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 2 | 0 | 3 | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Rash (Skin and subcutaneous tissue disorders) | 5 | 2 | 1 | 0 | 3 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 1 | NA | NA | NA
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Rash Pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Seborrhoeic Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Skin Irritation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Vitiligo (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Menopause (Social circumstances) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Arteriosclerosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Essential Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Hypertension (Vascular disorders) | 5 | 3 | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA
Orthostatic Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | 0 | NA | NA | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will with hold such publication for up to an additional 60 days to allow for filing of a patent application.

DOCUMENTS (2):
  • Study Protocol (2021-11-24): https://cdn.clinicaltrials.gov/large-docs/86/NCT03982186/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-19): https://cdn.clinicaltrials.gov/large-docs/86/NCT03982186/SAP_001.pdf